Replication of the P04334 Asthma Trial in Healthcare Claims Data

**DUPLICATE-P04334** 

September 14, 2021

NCT04892758

#### 1. RCT Details

This section provides a high-level overview of a **published** RCT that the described real-world evidence study is trying to replicate as closely as possible given the remaining limitations inherent in the healthcare databases.

#### 1.1 Title

Effects of Mometasone Furoate/Formoterol Combination Versus Mometasone Furoate Alone Versus Formoterol alone in Persistent Asthmatics (Study P04334AM1; NCT00383240)

#### 1.2 Intended aim(s)

To assess the effects of 26 weeks of treatment with mometasone furoate/formoterol (MF/F) compared with formoterol (F) alone on the incidence of time to first asthma deterioration in patients with persistent asthma previously receiving medium-dose inhaled corticosteroids.

# 1.3 Primary endpoint for replication

Asthma exacerbation defined by hospitalization or treatment with additional excluded asthma medication (i.e., systemic corticosteroids)

# 1.4 Required power for primary endpoint and noninferiority margin (if applicable)

This trial is a superiority trial. For time to first asthma deterioration, assuming a 5% event rate for MF/F 200/10 ug and an 18% event rate for F 10 ug, the trial's sample size will provide ~90% power to detect a treatment difference in survival curves.

#### 1.5 Trial estimate

The proportion of patients experiencing asthma deteriorations was MF/F, 30.4%, MF, 33.9%, F 54% (p <0.001). (Nathan et al., 2010). The calculated risk ratio is 0.90 (95% CI, 0.67-1.20) for MF/F vs MF and 0.56 (95% CI 0.44, 0.72) for MF/F vs F.

### 2. Person responsible for implementation of replication in Aetion

Hemin Lee, MD, MPH, implemented the study design in the Aetion Evidence Platform. She is not responsible for the validity of the design and analytic choices. All implementation steps are recorded, and the implementation history is archived in the platform.

# 3. Data Source(s)

Optum CDM, IBM® MarketScan®

# 4. Study Design Diagram

The study design diagram visualizes key aspects of the longitudinal study design for expedited review.

Figure 1. Design Diagram - P04334AM1 TRIAL REPLICATION

**Design Diagram - P04334 REPLICATION** Cohort Entry Date (Day 0) [Mometasone furoate/fomoterol fumarate OR 10 mcg fomoterol fumarate] INCL 1: Age ≥12 INCL 2: Utilization of medium daily dose of either ICS or ICS/LABA
Days [-180, 0] INCL 3: Recorded diagnosis of asthma Days [-365, 0] EXCL: Smoking or use of Nicotine Replacement Therapy EXCL: Oropharyngeal candidiasis [Days [-180, 0] PRIMARY OUTCOME(S): Covariate Assessment Window Days [-180, 0] Asthma Exacerbation Follow Up Window Days [1, censora] Time <sup>a</sup> Censoring criteria Day 0 Specified Date reached Occurrence of outcome Death Switch (within comparison grp) Start of additional Exposure • Nursing home admission End of index exposure

Disenrollment

#### 5. Cohort Identification

# 5.1 Cohort Summary

This study will involve a new user, parallel group, propensity score-matched, retrospective cohort design comparing mometasone-furoate/formoterol 200/10ug with formoterol 12 ug in patients with persistent asthma previously receiving medium-dose inhaled corticosteroids. The patients will be required to have continuous enrollment during a baseline period of 180 days before initiation of mometasone-furoate/formoterol or formoterol. (Note: the formoterol dose used in the trial was 10ug; in the replication, we will use the market available dose which is 12 ug).

### 5.2 <u>Important steps for cohort formation</u>

New use of mometasone-furoate/formoterol 200/10ug (exposure) is defined as no use of the exposure drug within the 180 days prior to index date. New use of formoterol 12 ug (comparator) is defined as no use of the comparator drug within the 180 days prior to index date. New users of mometasone-furoate/formoterol 200/10ug are not allowed to receive formoterol 12 ug within the 180 days prior to index date, and new users of formoterol 12 ug are not allowed to receive mometasone-furoate/formoterol 200/10ug within the 180 prior to index date.

#### 5.2.1 Eligible cohort entry dates

Mometasone-furoate/formoterol was approved by FDA on June 24, 2010 for the management of asthma. The initial eligible cohort entry date was the first date after June 24, 2010 for both the databases investigated (IBM® MarketScan®, Optum CDM). The last date eligible as cohort entry date was the end of available data for IBM® MarketScan® and Optum CDM. The following eligible cohort entry dates were included:

- Optum CDM: June 24, 2010 June 30, 2020 (end of available data)
- IBM® MarketScan®: June 24, 2010– December 31, 2018 (end of available data)
- 5.2.2 Specify <u>inclusion/exclusion</u> criteria for cohort entry and define the index date Inclusion and exclusion criteria were adapted from the trial as closely as possible. Definitions for all inclusion/exclusion are provided in **Appendix A** and are summarized in the flowcharts below.

## 5.3 Flowchart of the study cohort assembly

For Mometasone-furoate/formoterol vs. formoterol

| | Op | Optum | | etscan |
|---|---|---|---|---|
| Less Excluded Patients | Remaining<br>Patients | | Less Excluded Patients | Remaining<br>Patients |
| All patients | | 78,202,636 | | 200,203,908 |
| Did not meet cohort entry criteria | -<br>78,142,188 | 60,448 | 200,050,120 | 153,788 |
| Excluded due to insufficient enrollment | -8,307 | 52,141 | -16,744 | 137,044 |
| Excluded due to prior use of referent | -6,358 | 45,783 | -12,623 | 124,421 |
| Excluded due to prior use of exposure | -20,136 | 25,647 | -47,830 | 76,591 |
| Excluded because patient qualified in >1 exposure category | 0 | 25,647 | -4 | 76,587 |
| Excluded based on Age : Exclude missing | 0 | 25,647 | 0 | 76,587 |
| Excluded based on Gender: Exclude missing | 0 | 25,647 | 0 | 76,587 |
| Excluded based on INCLUSION: Age >=12 | -1,268 | 24,379 | -3,895 | 72,692 |
| Excluded based on Inclusion 3 - Medium dose ICS [-90,0] | -21,414 | 2,965 | -60,543 | 12,149 |
| Excluded based on Inclusion 4 - Asthma [-365, 0] | -587 | 2,378 | -1,947 | 10,202 |
| Excluded based on Inclusion 8 - Pregnancy | -7 | 2,371 | -14 | 10,188 |
| Excluded based on Exclusion 4/5 - Asthma exacerbation, respiratory failutre, Intubation [-90,0] | -890 | 1,481 | -1,153 | 9,035 |
| Excluded based on Exclusion 6 - Smoking | -63 | 1,418 | -112 | 8,923 |
| Excluded based on Exclusion 8 - Oropharyngeal candidiasis | -4 | 1,414 | -40 | 8,883 |
| Final cohort | | 1,414 | | 8,883 |

#### 6. Variables

## 6.1 Exposure-related variables:

#### Study drug:

New initiation of MF/F (200/10 ug twice daily). New initiation is defined as no use of MF/F in the prior 180 days before treatment initiation (washout period). New users of MF/F are not allowed to receive F within the 180 days prior to treatment initiation.

## Comparator agent:

New initiation of F (12 ug weekly). F 12ug is the market available dose form of formoterol that was selected for formoterol 10 ug used in the trial. New initiation is defined as no use of F in the prior 180 days before treatment initiation (washout period). New users of F are not allowed to receive MF/F 200/10 ug within the 180 days prior to treatment initiation.

## 6.2 Preliminary Covariates:

- Age
- Gender
- Combined Comorbidity Index (CCI), measured over the baseline covariate assessment period, defined as 180 days prior to and including index date.

Covariates listed above represent only a small subset of covariates that will ultimately be controlled for in the design and analysis. We use the covariates above only for initial feasibility analyses to judge whether there is likely to be sufficient overlap between treatment groups to proceed with the study. Remaining covariates are defined only after the study has passed the initial feasibility analysis and the initial power assessment and are listed in Table 1 (**Appendix B**).

# 6.3 Outcome variables and study follow-up:

#### 6.3.1 Outcome variables

Effectiveness outcome variables of interest (definitions provided in **Appendix A**):

- Primary outcome: Time to first asthma exacerbation (algorithm adapted from Nathan, et. al, and Fuhlbrigge A, et. al.,)
- 6.3.2 Study follow-up

Both as-treated (AT) and intention-to-treat (ITT) analyses will be conducted with treatment defined as the index drug on the day of cohort entry. Because adherence in the real-world databases is expected to be much worse than in the trial, the AT analysis is the primary analysis, as it targets the relative hazard of outcomes on treatment.

For the AT analyses, the follow-up will start the day after initiation of MF/F and F and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest,
- The date of end of continuous registration in the database,
- Discontinuation of the index drugs,
- End of the study period,
- Measured death event occurs,
- Nursing home admission
  - Nursing home admissions are considered a censoring event because the data sources utilized typically provide little to no data on a patient, particularly on drug utilization, after admission. We will utilize this as an exclusion reason for cohorts for the same reason.
- The date of drug discontinuation, defined as the date of the last continuous treatment episode of the index drug (MF/F and comparator) plus a defined grace period (i.e., 60 days after the end of the last prescription's days' supply in main analyses).
- The date of augmentation or switching from exposure to comparator or vice versa
  - A dosage change on the index treatment does not fulfill this criterion

### 7. Initial Feasibility Analysis

# Action report name:

For Mometasone-furoate/formoterol vs. formoterol

Optum CDM - https://bwh-dope.aetion.com/projects/details/1659/results/67130/result/0

IBM® MarketScan®- https://bwh-dope.aetion.com/projects/details/1658/results/66759/result/0

<u>Date conducted:</u> 03/07/2021 (Marketscan), 3/17/2021 (Optum)

Complete Aetion feasibility analysis using age and CCI as the only covariates and the primary endpoint (Section 6.3.1) as the outcome. No measures of association will be computed nor will incidence rates stratified by treatment group.

#### 8. Initial Power Assessment

## Aetion report name:

■ For Mometasone-furoate/formoterol vs. formoterol
Optum CDM - https://bwh-dope.aetion.com/projects/details/1659/results/67142/result/0
IBM® MarketScan®- https://bwh-dope.aetion.com/projects/details/1658/results/66760/result/0

Date conducted: 03/07/2021 (Marketscan), 3/17/2021 (Optum)

In order to complete the initial power analysis, the dummy outcome of a 90-day gap in database enrollment will be used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. Complete a 1:1 PS-matched comparative analysis using this outcome. PS should include only 3 covariates: age, gender, and combined comorbidity index. Power calculations are based on the formulas from Chow et al. (2008).

- Stop analyses until feasibility and power are reviewed by primary investigators and FDA. Reviewers evaluate the results of the analyses described above in Sections 7 and 8, including numbers of patients, patient characteristics, follow-up time, and reasons for censoring by treatment group, as well as overall rates of outcomes and study power. These parameters are re-evaluated and reported in the subsequent sections, after incorporating feedback and refining the protocol.
- Stop analyses until feasibility and power are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Shirley Wang | Date reviewed: | 3/19/2021 |
|-------------------------|--------------|----------------|-----------|
| Reviewed by FDA: | Ken Quinto | Date reviewed: | 4/2/2021 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

#### 9. Balance Assessment

For Mometasone-furoate/formoterol vs. formoterol

Optum CDM: https://bwh-dope.aetion.com/projects/details/1659/rwrs/68458 IBM® MarketScan®: https://bwh-dope.aetion.com/projects/details/1658/rwrs/68457

Date conducted:

04/14/2021

After review of initial feasibility and power analyses, complete creation of the remaining covariates from Section 6.2. Again, using the dummy outcome of a 90-day gap in database enrollment, complete a 1:1 PS-matched analysis. The PS should include the complete list of covariates.

- Provide plot of PS distributions stratified by treatment group. Note- Please refer to **Appendix B**.
- Report covariate balance after matching.

  Note- For Table 1, please refer to **Appendix B**.

Report reasons for censoring by treatment group.

| | Overall | Referent | Exposure |
|---|---|---|---|
| Dummy outcome | 0 (0.00%) | 0 (0.00%) | 0 (0.00%) |
| Death | 2 (0.09%) | 2 (0.09%) | 0 (0.00%) |
| Start of an additional exposure | 10 (0.46%) | 6 (0.28%) | 4 (0.18%) |
| End of index exposure | 1747 (80.58%) | 882 (40.68%) | 865 (39.90%) |
| Specified date reached | 4 (0.18%) | 0 (0.00%) | 4 (0.18%) |
| End of patient data | 0 (0.00%) | 0 (0.00%) | 0 (0.00%) |
| End of patient enrollment | 391 (18.04%) | 185 (8.53%) | 206 (9.50%) |
| Nursing home admission, pharmacy disenrollment | 14 (0.65%) | 9 (0.42%) | 5 (0.23%) |

• Report follow-up time by treatment group.

| Median Follow-Up Time (Days) [IQR] | | |
|---|---|---|
| Patient Group Optum Marketscan | | |
| Overall Patient Population | 133.5 [88,193] | 141.5 [88,214] |
| Referent | 123 [88,157] | 147 [88, 207] |
| Exposure | 138 [88,254] | 132 [88,222] |

• Report overall risk of the primary outcome.

Effectiveness research with Real World Data to support FDA's regulatory decision making

| | Optum CDM | IBM® MarketScan® | Pooled |
|-------------------------|-----------|------------------|--------|
| Risk per 1,000 patients | 125.88 | 144.24 | 141.6 |

## 10. Final Power Assessment

Date conducted: 4/15/2021

• Re-calculate power in the appropriate excel table, using the revised number of matched patients from the PS-match in Section 9. All other parameters in the table should be the same as in Section 8.

o <u>Pooled</u>

| Superiority Analysis | |
|----------------------------|----------|
| Number of patients matched | 2,168 |
| Reference | 1,084 |
| Exposed | 1,084 |
| Risk per 1,000 patients | 141.60 |
| Desired HR from RCT | 0.28 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 306.9888 |
| Power | 1 |

Optum CDM

| Superiority Analysis | |
|----------------------------|------------|
| Number of patients matched | 330 |
| Reference | 165 |
| Exposed | 165 |
| Risk per 1,000 patients | 125.88 |
| Desired HR from RCT | 0.28 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 41.5404 |
| Power | 0.98391473 |

o <u>IBM® MarketScan®</u>

| 1,838 |
|-----------|
| 919 |
| 919 |
| 144.24 |
| 0.28 |
| 0.05 |
| 265.11312 |
| 1 |

• Stop analyses until balance and final power assessment are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Shirley Wang | Date reviewed: | 4/16/2021 |
|-------------------------|--------------|----------------|-----------|
| Reviewed by FDA: | Ken Quinto | Date reviewed: | 4/30/2021 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

# 11. Study Confidence and Concerns

<u>Deadline for voting on study confidence and listing concerns:</u> <u>Date votes and concerns are summarized:</u>

- If final feasibility and power analyses are reviewed and approved, proceed to the remaining protocol steps.
- All study team and advisory board members that review this protocol should at this stage provide their level of confidence for the
  success of the RWD study in the <u>Google Form</u>. This form also provides space for reviewers to list any concerns that they feel may
  contribute to a failure to replicate the findings of the RCT, including differences in study populations, poor measurement of study
  variables, or residual confounding. All responses will be kept confidential and individual-level results will only be shared with the
  individual respondent.
- After the deadline for voting has passed, provide the distribution of responses and summarize all concerns here.

# 12. Register study protocol on clinicalTrials.gov

Date conducted:

• Register the study on <u>clinicalTrials.gov</u> and upload this document.

#### 13. Comparative Analyses

Action report name:

Date conducted:

# 13.1 For primary analysis:

# 13.2 For sensitivity analyses:

# 14. Requested Results

# 14.1 <u>Table 1: Baseline characteristics before and after adjustment</u>

| Variable | Before adjustment | | After adjustment | | | |
|---|---|---|---|---|---|---|
| | Referent | Exposure | Std. diff. | Referent | Exposure | Std. diff. |
| Number of patients | | | - | | | - |
| Age categories | | | | | | |

# 14.2 <u>Table 2: Follow-up time</u>

| Patient Group | Median Follow-Up Time (Days) [IQR] |
|----------------------------|------------------------------------|
| Overall Patient Population | |
| Referent | |
| Exposure | |

# 14.3 <u>Table 3: Censoring events</u>

| | Overall | Referent | Exposure |
|---|---|---|---|
| Dummy outcome | | | |
| Death | | | |
| Start of an additional exposure | | | |
| End of index exposure | | | |
| Specified date reached | | | |
| End of patient data | | | |
| End of patient enrollment | | | |
| Nursing home admission, pharmacy disenrollment | | | |

## 14.4 Table 4: Results from primary analyses;

| Analysis | No. exposed events | No. referent events | Exposed rate | Referent rate | HR (95% CI) |
|---|---|---|---|---|---|
| Crude | | | | | |
| Analysis 1 | | | | | |
| Analysis 2 | | | | | |

HR, Hazard Ratio; CI, Confidence Interval.

# 14.5 <u>Table 5: Results from secondary analyses.</u>

## 15. References

Fuhlbrigge A, Peden D, Apter AJ, et al. Asthma outcomes: exacerbations. *J Allergy Clin Immunol*. 2012;129(3 Suppl):S34-S48. doi:10.1016/j.jaci.2011.12.983

Nathan RA, Nolte H, Pearlman DS; P04334 Study Investigators. Twenty-six-week efficacy and safety study of mometasone furoate/formoterol 200/10 microg combination treatment in patients with persistent asthma previously receiving medium-dose inhaled corticosteroids. Allergy Asthma Proc. 2010 Jul-Aug;31(4):269-79. doi: 10.2500/aap.2010.31.3364. Epub 2010 Jul 30. PMID: 20678306.

Chow S, Shao J, Wang H. 2008. *Sample Size Calculations in Clinical Research*. 2nd Ed. Chapman & Hall/CRC Biostatistics Series. page 177.

| # | P04334AM1 trial definitions | Implementation in routine care | Please see the following Google Drive for further details or<br>https://drive.google.com/drive/folders/1WD618wrywYEaXdLTd | | Color Coding Criteria Can be replicated in claims |
|---|---|---|---|---|---|
| | Trial details- clinicaltrials.gov N<br>EXPOSURE vs. COMPAF | | ICD-10 codes are not listed in this document because of excel cell size ICD-10 codes. Full ICD-10 code lists will be available in the above Goog ICD-10 codes coversions were completed using a 5A5 macro that implication in the code of the CMS ICD-9 to ICD-10 map https://www.nbe.org/data/rcd3-icd-10-mand-ocs-crosswalk-sea | limitations and excessive number of gle Drive Folder (link above). ICD-9 to lements forward/ backward mapping oping: | Using dummy definitions for measuring in claims Can't be measured in claims Can't be measured in claims but not important for the analysis |
| | Exposure ) Mometasone furoate/formoterol fumarate combination MDI 200/10 mcg BID vs.<br>Referent) Formoterol fumarate 10 mcg | Exposure: Mometasone furoate/formoterol fumarate 200/10 mcg BID NDC.code: 00085720601 00085720607 Referent: formoterol fumarate 10 mcg NDC.code: 54599575400 - formoterol fumarate 54568497200 - formoterol fumarate 54686497200 - formoterol fumarate 50083016702 - formoterol fumarate 00083016701 - formoterol fumarate 00083016701 - formoterol fumarate 00083016701 - formoterol fumarate 00083016701 - formoterol fumarate 00083016701 - formoterol fumarate 00085140201 - formoterol fumarate 00085140201 - formoterol fumarate 60085140201 - formoterol fumarate 68115065160 - formoterol fumarate 68115065160 - formoterol fumarate | | | |
| | PRIMARY OUTCOM Time-to-first Asthma Exacerbation | Measured 1 day after drug initiation 1) Asthma diagnosis code in inpatient primary diagnosis position 2) Asthma diagnosis code in inpatient any position or outpatient setting PLUS a prescription claim for systemic steroids 14 days before and after the diagnosis code Asthma: ICD-9: 493.x ICD-10: 145.* | | | |
| | INCLUSION CRITERI | | | | |
| 3 | Informed Consent: A signed and dated written informed consent prior to study participation Age ≥ 12 years, adult and adolescent subjects A subject must have been using a medium daily dose of inhaled glucocorticosteroid (ICS) (either alone or in combination with a long-acting beta agonist (LABA)) for at least 12 weeks and must have been on a stable regimen (daily dose unchanged) for at least 2 weeks prior to Screening. Medium daily doses of ICS are defined as follows: 5500 to 1000 mcg beclomethasone chlorofluorocarbon (CFC) 2500 to 500 mcg beclomethasone hydrofluoroalikane (HFA) 5600 to 1000 mcg budesonide dry powder inhaler (DPI) 2500 to 500 mcg fluitsolide 250 to 500 mcg fluitcasone 400 mcg MF 21000 to 2000 mcg triamcinolone acetonide | N/A Measured on the day of drug of initiation Age >= 12 Measured 90 days prior to drug initiation See tab [medium dose ICS] for NDC codes | | | |
| 4 | To document the diagnosis of asthma and assure the subject's responsiveness to bronchodilators before randomization one of the following methods can be used at the Screening Visit, Day -14, or thereafter, but prior to the Baseline Visit: The subject must demonstrate an increase in absolute FEV1 of at least 12% and at least 200 mL within 15 minutes after administration of four inhalations of albuterol/salbutamol (total dose of 360 to 400 mgg) or of nebulized SABA (2.5 mg) if confirmed as standard office practice, OR The subject must demonstrate a peak expiratory flow (PEF) variability of more than 20% expressed as a percentage of the highest and lowest morning prebronchodilator PEF over at least 1 week OR The subject must demonstrate a diurnal variation in PEF of more than 20% based on the difference between the prebronchodilator morning value and the postbronchodilator value from the evening before, expressed as a percentage of the mean daily PEF value. | Measured 365 days prior to cohort entry in any position, any setting Asthma: ICD-9: 493.x ICD-10: J45.* | Larsson K, Ställberg B, Lisspers K, Telg G, Johansson G, Thuresson M,<br>Janson C, Prevalence and management of severe asthma in primary<br>care: an observational cohort study in Swedner (PACEH), Respir Res.<br>2018 Jan 18:19(1):12. doi: 10.1186/s12931-018-0719-x. PMID:<br>29347939; PMCID: PMC5774144. | | |
| 5 6 | At the Screening Visit, the subject's FEV1 must be ≥60% and ≤90% predicted. At the Baseline Visit, the subject's FEV1 must be ≥60% and ≤85% predicted when all restricted medications have been withheld for the appropriate intervals. Clinical laboratory tests (complete blood counts [CBC], blood chemistries, and urinalysis) conducted at the Screening Visit must be within normal limits or clinically acceptable to the investigator/sponsor. An electrocardiogram (ECG) using a centralized trans-telephonic technology at the Screening Visit must be clinically acceptable to the investigator. A chest-vray performed at the Screening Visit, or within 12 months prior to the Screening Visit, must be clinically acceptable to the investigator. | N/A<br>N/A | | | |

# Appendix A

| 8 | A female subject of childbearing potential must have been using a medically acceptable, adequate form of birth control. This includes: 1) hormonal contraceptives as prescribed by a physician (oral combined, hormonal implant); 2) medically prescribed intra-uterine device (IUD); 3) condom in combination with a spermicide (double barrier method); 4) monogamous relationship with a male partner who has had a vasectomy. The subject must have started this birth control method at least 3 months prior to Screening (with the exception of condom in combination with spermicide), and must agree to continue its use for the duration of the study. A female subject of childbearing potential who is not currently sexually active must agree and consent to using a medically acceptable birth control method should she become sexually active during the course of this study. Women who have been surgicially sterilized or are at least 1 year postmenopaula are not considered to be of childbearing potential. A female subject of childbearing potential must have a negative serum pregnancy test at Screening in order to be considered eligible for enrollment. EXCLUSION CRITER | Measured 180 days prior to drug initiation in any setting and position See tab [pregnancy]; will be applied as an exclusion. | |
|---|---|---|---|
| | A subject who demonstrates a change (increase or decrease) in absolute FEV1 of >20% at any time from the | N/A | |
| 1 | Screening Visit up to and including the Baseline Visit. | 77. | |
| 2 | A subject who requires the use of greater than eight inhalations per day of SABA MDI, or two or more nebulized treatments per day of 2.5 mg SABA, on any 2 consecutive days from the Screening Visit up to and including the Baseline Visit. | N/A | |
| 3 | A subject who experiences a decrease in AM or PM PEF below the Screening Period stability limit on any 2 consecutive days prior to Randomization. | N/A | |
| | | Measured 90 days prior to drug initiation | |
| 4 | A subject who experiences an occurrence of any clinical deterioration of asthma that results in emergency<br>treatment, hospitalization due to asthma, or treatment with additional, excluded asthma medication (other<br>than SABA) as judged by the clinical investigator at any time from the Screening Visit up to and including the<br>Baseline Visit. | Asthma exacerbation 1) Asthma diagnosis code in inpatient primary diagnosis position 2) Asthma diagnosis code in inpatient any position or outpatient setting PLUS a prescription claim for systemic steroids 14 days before and after the diagnosis code | |
| 5 | Emergency room treatment for asthma deterioration requiring systemic corticosteroid therapy or hospitalization for managemenet of airway obstruction within the 3 months before baseline | Asthma: (CD-9: 493.x) (CD-10: 145.*) or Acute respiratory failure/insufficiency/arrest (CD-9: 517.3", "518.5", "518.81", "518.82", "518.84", "799.1", "V46.1", "V46.11", "V46.12", "V46.13", "V46.2", "196.10", "196.11", "196.12", "196.20", "196.22", "196.20", "196.01", "196.02", "196.11", "196.12", "196.22", "196.22", "196.22", "196.90", "196.92", "R09.01", "R09.2", "299.11", "299.12", "299.81" } Intubation/Non-invasive ventilatory support: (CD-9 Procedure code: "03.90", "93.92", "96.01", "96.02", "96.03", "96.04", "96.05", "96.70", "96.71", "96.72", "96.72", "09.11", "96.72", "09.11722", "09.11822", "06.17722", "0CH/882", "00H/5722", "09H/582", "0WHQ722", "0WHQ722", "5A09357", "5A09457", "5A09557", "5A19352", "5A19452", "5A19552" } | Walkey AJ, Wiener RS. Use of noninvasive ventilation in patients with acute respiratory failure, 2000-2009: a population-based study. Ann Am Thoras Sc. 2013 Reb. 10(1):107. doi: 10.1513/AnnalsATS.201206-034OC. PMID: 23509327; PMCID: PMC3780971. |
| 6 7 | A subject who is a smoker or ex-smoker and has smoked within the previous year or has had a cumulative smoking history >10 pack-years Patients requiring concomitant asthma medication Clinically significant abnormal vital sign | Measured 180 days prior to drug initiation in any setting, any position ICD-9/10 codes: V15.82, 305.1x, 649.0x, 989.84 OR CPT code 99406, 99407, G0436, G0437, G9016, S9075, S9453, S4995, G9276, G9458, 1034F, 4004F, 4001F OR use of varenicline tartrate or nicotine replacement therapy ("Nicotine", "Nicotine Bitartrate", and "Nicotine Polacrilex") N/A N/A Measured 180 days prior to drug initiation in any setting, any position | |
| 8 | Visible evidence of oropharyngeal candidiasis at baseline or earlier | <u>Oropharyngeal candidiasis:</u><br>ICD-9: 112.0<br>ICD-10: B37.0, B37.83 | |

| NDC codes for medium dose ICS |
|-------------------------------|
| 37024523 |
| 85134107 |
| 85433401 |
| 85461001 |
| 173049500 |
| 173050400 |
| 173060100 |
| 173060102 |
| 173069604 |
| 173071700 |
| 173071722 |
| 173072000 |
| 173072020 |
| 173075300 |
| 173085914 |
| 173087414 |
| 173088710 |
| 173088714 |
| 21695019601 |
| 23490754201 |
| 35356009914 |
| 49999061412 |
| 49999081960 |
| 54569524200 |
| 54569566300 |
| 54868554700 |
| 54868563700 |
| 55045335400 |
| 58016481201 |
| 59310071106 |
| 68115092460 |
| 68258303101 |
| 85134101 |
| 85134102 |

| 85134103 |
|-------------|
| 85134104 |
| 85134106 |
| 85461005 |
| 93360982 |
| 173049900 |
| 173060202 |
| 173069600 |
| 173069602 |
| 173071720 |
| 173085910 |
| 173088810 |
| 49999061401 |
| 54569460200 |
| 54569460300 |
| 54569570200 |
| 54868439200 |
| 54868451700 |
| 54868554701 |
| 54868554702 |
| 55045291901 |
| 55045368601 |
| 58016460401 |
| 59310072206 |
| 59310082206 |
| 68115063713 |
| 68258891306 |

72.52 OTHER PARTIAL BREECH EXTRACTION

# Pregnancy Diagnosis codes 650 NORMAL DELIVERY 660 OBSTRUCTED LABOR 661 ABNORMALITY OF FORCES OF LABOR 662 LONG LABOR 663 UMBILICAL CORD COMPLICATIONS DURING LABOR AND DELIVERY 664 TRAUMA TO PERINEUM AND VULVA DURING DELIVERY 665 OTHER OBSTETRICAL TRAUMA 667 RETAINED PLACENTA OR MEMBRANES WITHOUT HEMORRHAGE 668 COMPLICATIONS OF THE ADMINISTRATION OF ANESTHETIC OR OTHER SEDATION IN LABOR AND DELIVERY 669.94 UNSPECIFIED COMPLICATION OF LABOR AND DELIVERY POSTPARTUM CONDITION OR COMPLICATION V24 POSTPARTUM CARE AND EXAMINATION V24.0 POSTPARTUM CARE AND EXAMINATION IMMEDIATELY AFTER DELIVERY V24.1 POSTPARTUM CARE AND EXAMINATION OF LACTATING MOTHER V24.2 ROUTINE POSTPARTUM FOLLOW V27 OUTCOME OF DELIVERY V27.0 MOTHER WITH SINGLE LIVEBORN V27.1 MOTHER WITH SINGLE STILLBORN+A2:J81 V27.2 MOTHER WITH TWINS BOTH LIVEBORN V27.3 MOTHER WITH TWINS ONE LIVEBORN AND ONE STILLBORN V27.4 MOTHER WITH TWINS BOTH STILLBORN V27.5 MOTHER WITH OTHER MULTIPLE BIRTH ALL LIVEBORN V27.6 MOTHER WITH OTHER MULTIPLE BIRTH SOME LIVEBORN V27.7 MOTHER WITH OTHER MULTIPLE BIRTH ALL STILLBORN V27.9 MOTHER WITH UNSPECIFIED OUTCOME OF DELIVERY Procedure codes 72.0 LOW FORCEPS OPERATION 72.1 LOW FORCEPS OPERATION WITH EPISIOTOMY 72.2 MID FORCEPS OPERATION 72.21 MID FORCEPS OPERATION WITH EPISIOTOMY 72.29 OTHER MID FORCEPS OPERATION 72.3 HIGH FORCEPS OPERATION 72.31 HIGH FORCEPS OPERATION WITH EPISIOTOMY 72.39 OTHER HIGH FORCEPS OPERATION 72.4 FORCEPS ROTATION OF FETAL HEAD 72.5 BREECH EXTRACTION 72.51 PARTIAL BREECH EXTRACTION WITH FORCEPS TO AFTERCOMING HEAD

## Appendix A

- 72.53 TOTAL BREECH EXTRACTION WITH FORCEPS TO AFTERCOMING HEAD
- 72.54 OTHER TOTAL BREECH EXTRACTION
- 72.6 FORCEPS APPLICATION TO AFTERCOMING HEAD
- 72.7 VACUUM EXTRACTION
- 72.71 VACUUM EXTRACTION WITH EPISIOTOMY
- 72.79 OTHER VACUUM EXTRACTION
- 72.8 OTHER SPECIFIED INSTRUMENTAL DELIVERY
- 72.9 UNSPECIFIED INSTRUMENTAL DELIVERY
- 73.0 ARTIFICIAL RUPTURE OF MEMBRANES
- 73.01 INDUCTION OF LABOR BY ARTIFICIAL RUPTURE OF MEMBRANES
- 73.09 OTHER ARTIFICIAL RUPTURE OF MEMBRANES
- 73.1 OTHER SURGICAL INDUCTION OF LABOR
- 73.2 INTERNAL AND COMBINED VERSION AND EXTRACTION
- 73.21 INTERNAL AND COMBINED VERSION WITHOUT EXTRACTION
- 73.22 INTERNAL AND COMBINED VERSION WITH EXTRACTION
- 73.3 FAILED FORCEPS
- 73.4 MEDICAL INDUCTION OF LABOR
- 73.5 MANUALLY ASSISTED DELIVERY
- 73.51 MANUAL ROTATION OF FETAL HEAD
- 73.59 OTHER MANUALLY ASSISTED DELIVERY
- 73.6 EPISIOTOMY
- 73.8 OPERATIONS ON FETUS TO FACILITATE DELIVERY
- 73.9 OTHER OPERATIONS ASSISTING DELIVERY
- 73.91 EXTERNAL VERSION ASSISTING DELIVERY
- 73.92 REPLACEMENT OF PROLAPSED UMBILICAL CORD
- 73.93 INCISION OF CERVIX TO ASSIST DELIVERY
- 73.94 PUBIOTOMY TO ASSIST DELIVERY
- 73.99 OTHER OPERATIONS ASSISTING DELIVERY
- 74.0 CLASSICAL CESAREAN SECTION
- 74.1 LOW CERVICAL CESAREAN SECTION
- 74.2 EXTRAPERITONEAL CESAREAN SECTION
- 74.3 REMOVAL OF EXTRATUBAL ECTOPIC PREGNANCY
- 74.4 CESAREAN SECTION OF OTHER SPECIFIED TYPE
- 74.9 CESAREAN SECTION OF UNSPECIFIED TYPE
- 74.91 HYSTEROTOMY TO TERMINATE PREGNANCY
- 74.99 OTHER CESAREAN SECTION OF UNSPECIFIED TYPE
- 75.4 MANUAL REMOVAL OF RETAINED PLACENTA
- 75.5 REPAIR OF CURRENT OBSTETRIC LACERATION OF UTERUS
- 75.6 REPAIR OF OTHER CURRENT OBSTETRIC LACERATION
- 75.7 MANUAL EXPLORATION OF UTERINE CAVITY, POSTPARTUM
- 75.9 OTHER OBSTETRIC OPERATIONS



| | Unmatched | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Opti | ım | | Mai | rketscan | | PC | OOLED | |
| | Formoterol fumarate | Mometasone | • | Formoterol fumarate | Mometasone | | Formoterol fumarate | Mometasone | |
| Variable | 10 mcg | furoate/formoterol | St. Diff. | 10 mcg | furoate/formoterol | St. Diff. | 10 mcg | furoate/formoterol | St. Diff. |
| North an of making the | | fumarate | | , and the second | fumarate | | ū | fumarate | |
| Number of patients | 363 | 1,051 | | 1,325 | 7,549 | | 1,688 | 8,600 | ' |
| Year of Cohort Entry Date | 70 (24 50/) | 7 (0.7%) | 0.063 | 205 (22 09/) | 112 /1 50/ | 0.061 | 202 (22 70/) | 110 (1 40/) | 0.692 |
| 2010; n (%) | 78 (21.5%) | , , | 0.062 | 305 (23.0%) | 112 (1.5%) | | 383 (22.7%) | 119 (1.4%) | |
| 2011; n (%) | 115 (31.7%) | 121 (11.5%) | 0.044 | 385 (29.1%) | 992 (13.1%) | 0.035 | 500 (29.6%) | 1,113 (12.9%) | 0.417 |
| 2012; n (%) | 67 (18.5%) | 173 (16.5%) | 0.005 | 258 (19.5%) | 1,275 (16.9%) | 0.006 | 325 (19.3%) | 1,448 (16.8%) | 0.065 |
| 2013; n (%) | 41 (11.3%) | 174 (16.6%) | -0.014 | 143 (10.8%) | 1,173 (15.5%) | -0.013 | 184 (10.9%) | 1,347 (15.7%) | -0.142 |
| 2014; n (%) | 37 (10.2%) | 163 (15.5%) | -0.015 | 142 (10.7%) | 1,700 (22.5%) | -0.029 | 179 (10.6%) | 1,863 (21.7%) | -0.305 |
| 2015; n (%) | 20 (5.5%) | 142 (13.5%) | -0.026 | 79 (6.0%) | 846 (11.2%) | -0.018 | 099 (5.9%) | 988 (11.5%) | -0.200 |
| 2016; n (%) | 5 (1.4%) | 124 (11.8%) | -0.041 | 13 (1.0%) | 679 (9.0%) | -0.036 | 018 (1.1%) | 803 (9.3%) | -0.376 |
| 2017; n (%) | 0 (0.0%) | 59 (5.6%) | -0.033 | 0 (0.0%) | 500 (6.6%) | -0.036 | 000 (0.0%) | 559 (6.5%) | -0.373 |
| 2018; n (%) | 0 (0.0%) | 30 (2.9%) | -0.024 | 0 (0.0%) | 272 (3.6%) | -0.027 | 000 (0.0%) | 302 (3.5%) | -0.269 |
| 2019; n (%) | 0 (0.0%) | 34 (3.2%) | -0.025<br>-0.021 | NA<br>NA | NA<br>NA | NA | NA<br>NA | NA<br>NA | NA<br>NA |
| 2020; n (%) | 0 (0.0%) | 24 (2.3%) | -0.021 | NA | NA | NA | NA | NA | INA |
| Age | 55.06 (45.04) | 50.76 (47.04) | 0.271 | FC F7 (1F OC) | 46 67 (10 21) | 0.580 | FC 30 /4 F 7F) | 47 17 (10 16) | 0.537 |
| mean (sd) | 55.26 (15.34) | 50.76 (17.81) | 0.271 | 56.57 (15.86)<br>59.00 [48.00, 65.00] | 46.67 (18.21) | 0.580 | 56.29 (15.75) | 47.17 (18.16) | 0.537 |
| median [IQR] | 57.00 [48.00, 65.00] | 53.00 [40.00, 63.00] | 0.241 | J3.UU [46.UU, 65.UU] | 50.00 [34.00, 60.00] | 0.527 | 58.57 (15.75) | 50.37 (18.16) | 0.482 |
| Age categories12-17; n (%) | 11 (3.0%) | 68 (6.5%) | -0.016 | 35 (2.6%) | 800 (10.6%) | -0.031 | 046 (2.7%) | 868 (10.1%) | -0.306 |
| | | | | | | -0.031 | | | -0.308 |
| 18-39; n (%) | 39 (10.7%) | 182 (17.3%) | -0.018 | 124 (9.4%) | 1,588 (21.0%) | | 163 (9.7%) | 1,770 (20.6%) | |
| 40 - 64; n (%) | 221 (60.9%) | 574 (54.6%) | 0.008 | 814 (61.4%) | 4,178 (55.3%) | 0.008<br>0.031 | 1,035 (61.3%) | 4,752 (55.3%) | 0.122<br>0.307 |
| >= 65; n (%) | 92 (25.3%) | 227 (21.6%) | 0.008 | 352 (26.6%) | 983 (13.0%) | 0.031 | 444 (26.3%) | 1,210 (14.1%) | 0.307 |
| Geographic Region | 46 (12 70/) | 97 (9.2%) | 0.011 | 332 (25.1%) | 1 220 /16 49/\ | 0.019 | 270 (22 40/) | 1 226 /15 50/\ | 0.177 |
| Northeast; n (%) | 46 (12.7%) | 392 (37.3%) | | 447 (33.7%) | 1,239 (16.4%) | | 378 (22.4%) | 1,336 (15.5%) | 0.177 |
| South; n (%) | 163 (44.9%) | 392 (37.3%)<br>372 (35.4%) | 0.012<br>-0.022 | , , | 2,643 (35.0%) | -0.002 | 610 (36.1%) | 3,035 (35.3%) | 0.017 |
| Midwest; n (%) | 86 (23.7%) | 190 (18.1%) | 0.022 | 307 (23.2%) | 1,605 (21.3%) | 0.004<br>-0.020 | 393 (23.3%) | 1,977 (23.0%) | |
| West; n (%) | 68 (18.7%) | 190 (18.1%)<br>NA | NA | 222 (16.8%)<br>17 (1.3%) | 1,972 (26.1%)<br>90 (1.2%) | 0.020 | 290 (17.2%) | 2,162 (25.1%)<br>NA | -0.194<br>NA |
| Unknown/Missing; n (%) Metropolitan Statistical Area | NA | INA | INA | 17 (1.5%) | 90 (1.2%) | 0.001 | NA | NA | INA |
| • | NA | NA | NA | 1,090 (82.3%) | 6,106 (80.9%) | 0.002 | NA | NA | NA |
| Urban; n (%)<br>Rural; n (%) | NA<br>NA | NA<br>NA | NA | 2 (0.2%) | 132 (1.7%) | -0.015 | NA<br>NA | NA<br>NA | NA |
| Unknown/Missing; n (%) | NA<br>NA | NA<br>NA | NA | 233 (17.6%) | 1,311 (17.4%) | 0.000 | NA<br>NA | NA<br>NA | NA |
| General Health Related Measures | INA | INA | IVA | 233 (17.0%) | 1,311 (17.4%) | 0.000 | IVA | INA | INA |
| Alcohol/Drug abuse or dependence ; n (%) | 6 (1.7%) | 23 (2.2%) | -0.004 | 18 (1.4%) | 76 (1.0%) | 0.004 | 024 (1.4%) | 099 (1.2%) | 0.018 |
| Obesity or Overweight; n (%) | 39 (10.7%) | 133 (12.7%) | -0.004 | 104 (7.8%) | 694 (9.2%) | -0.005 | 143 (8.5%) | 827 (9.6%) | -0.038 |
| Obesity; n (%) | 35 (9.6%) | 109 (10.4%) | -0.003 | 93 (7.0%) | 594 (7.9%) | -0.003 | 128 (7.6%) | 703 (8.2%) | -0.038 |
| Overweight; n (%) | 4 (1.1%) | 27 (2.6%) | -0.003 | 14 (1.1%) | 112 (1.5%) | -0.003 | 018 (1.1%) | 139 (1.6%) | -0.022 |
| Cardiovascular Measures | 4 (1.170) | 27 (2.070) | -0.011 | 14 (1.170) | 112 (1.570) | -0.004 | 010 (1.170) | 133 (1.0%) | -0.043 |
| Hypertension; n (%) | 165 (45.5%) | 403 (38.3%) | 0.011 | 537 (40.5%) | 2,096 (27.8%) | 0.022 | 702 (41.6%) | 2,499 (29.1%) | 0.264 |
| Hyperlipidemia; n (%) | 135 (37.2%) | 320 (30.4%) | 0.012 | 419 (31.6%) | 1,621 (21.5%) | 0.022 | 554 (32.8%) | 1,941 (22.6%) | 0.229 |
| MI, angina, Coronary atherosclerosis and other forms of chronic | 155 (57.270) | 320 (30.470) | 0.012 | 413 (31.0%) | 1,021 (21.570) | 0.020 | 334 (32.0%) | 1,541 (22.070) | 0.223 |
| ischemic heart disease; n (%) | 39 (10.7%) | 56 (5.3%) | 0.019 | 159 (12.0%) | 300 (4.0%) | 0.028 | 198 (11.7%) | 356 (4.1%) | 0.285 |
| Old MI; n (%) | 6 (1.7%) | 7 (0.7%) | 0.009 | 12 (0.9%) | 20 (0.3%) | 0.008 | 018 (1.1%) | 027 (0.3%) | 0.096 |
| Acute MI; n (%) | 2 (0.6%) | 3 (0.3%) | 0.004 | 8 (0.6%) | 10 (0.1%) | 0.008 | 010 (0.6%) | 013 (0.2%) | 0.063 |
| Stable angina; n (%) | 5 (1.4%) | 5 (0.5%) | 0.009 | 16 (1.2%) | 47 (0.6%) | 0.006 | 021 (1.2%) | 052 (0.6%) | 0.064 |
| Coronary atherosclerosis and other forms of chronic ischemic | 3 (2.770) | 5 (5.570) | | | | | | | |
| heart disease; n (%) | 36 (9.9%) | 52 (4.9%) | 0.018 | 143 (10.8%) | 252 (3.3%) | 0.028 | 179 (10.6%) | 304 (3.5%) | 0.280 |
| History of CABG or PTCA; n (%) | 4 (1.1%) | 11 (1.0%) | 0.001 | 14 (1.1%) | 28 (0.4%) | 0.008 | 018 (1.1%) | 039 (0.5%) | 0.067 |
| Cerebrovascular disease (Stroke, TIA, Late effects); n (%) | 7 (1.9%) | 16 (1.5%) | 0.003 | 21 (1.6%) | 62 (0.8%) | 0.007 | 028 (1.7%) | 078 (0.9%) | 0.071 |
| Stroke (Ischemic or hemorrhagic); n (%) | 7 (1.9%) | 8 (0.8%) | 0.009 | 13 (1.0%) | 31 (0.4%) | 0.007 | 020 (1.2%) | 039 (0.5%) | 0.076 |
| TIA; n (%) | 0 (0.0%) | 8 (0.8%) | -0.013 | 10 (0.8%) | 24 (0.3%) | 0.007 | 010 (0.6%) | 032 (0.4%) | 0.028 |
| Late effects of cerebrovascular disease; n (%) | 2 (0.6%) | 4 (0.4%) | 0.003 | 7 (0.5%) | 19 (0.3%) | 0.003 | 009 (0.5%) | 023 (0.3%) | 0.032 |
| Atrial fibrillation and Other cardiac dysrhythmia; n (%) | 25 (6.9%) | 75 (7.1%) | -0.001 | 108 (8.2%) | 320 (4.2%) | 0.016 | 133 (7.9%) | 395 (4.6%) | 0.137 |
| Atrial fibrillation; n (%) | 10 (2.8%) | 40 (3.8%) | -0.006 | 64 (4.8%) | 150 (2.0%) | 0.015 | 074 (4.4%) | 190 (2.2%) | 0.123 |
| Other cardiac dysrhythmia; n (%) | 20 (5.5%) | 59 (5.6%) | 0.000 | 65 (4.9%) | 231 (3.1%) | 0.009 | 085 (5.0%) | 290 (3.4%) | 0.080 |
| Diabetes Related Measures | ( | () | | • • | , , | | , , | , , | |
| Diabetes with or w/o complications; n (%) | 52 (14.3%) | 155 (14.7%) | -0.001 | 227 (17.1%) | 706 (9.4%) | 0.021 | 279 (16.5%) | 861 (10.0%) | 0.193 |
| | | \ | | | | | | | |

| | • | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Diabetes mellitus without mention of complications; n (%) | 50 (13.8%) | 149 (14.2%) | -0.001 | 214 (16.2%) | 670 (8.9%) | 0.021 | 264 (15.6%) | 819 (9.5%) | 0.185 |
| Diabetes with specified complications; n (%) | 9 (2.5%) | 40 (3.8%) | -0.007 | 52 (3.9%) | 119 (1.6%) | 0.014 | 061 (3.6%) | 159 (1.8%) | 0.111 |
| Diabetes with unspecified complications; n (%) | 2 (0.6%) | 4 (0.4%) | 0.003 | 10 (0.8%) | 24 (0.3%) | 0.007 | 012 (0.7%) | 028 (0.3%) | 0.057 |
| GI Conditions | | | 0.007 | 474 (42 000) | 4.044(40.40() | 0.004 | 220 (42 50() | 4 200 (4 4 40() | 0.047 |
| GERD; n (%) | 57 (15.7%) | 195 (18.6%) | -0.007 | 171 (12.9%) | 1,014 (13.4%) | -0.001 | 228 (13.5%) | 1,209 (14.1%) | -0.017 |
| Upper GI (Diseases of esophagus, stomach and duodenum including GERD); n (%) | CO (40 70/) | 247 (20 (0/) | -0.004 | 222 (16.8%) | 1,216 (16.1%) | 0.002 | 290 (17.2%) | 1,433 (16.7%) | 0.013 |
| GI bleeding; n (%) | 68 (18.7%) | 217 (20.6%) | 0.009 | 21 (1.6%) | 85 (1.1%) | 0.004 | 030 (1.8%) | 099 (1.2%) | 0.049 |
| Non-infective enteritis and colitis; n (%) | 9 (2.5%)<br>13 (3.6%) | 14 (1.3%)<br>49 (4.7%) | -0.005 | 62 (4.7%) | 257 (3.4%) | 0.004 | 075 (4.4%) | 306 (3.6%) | 0.049 |
| Intraoperative and postprocedural complications and disorders of | | | | | | | | | |
| digestive system; n (%) | 10 (2.8%) | 16 (1.5%) | 0.009 | 26 (2.0%) | 106 (1.4%) | 0.005 | 036 (2.1%) | 122 (1.4%) | 0.053 |
| Disorders of gallbladder, biliary tract and pancreas; n (%) | 1 (0.3%) | 18 (1.7%) | -0.014 | 15 (1.1%) | 82 (1.1%) | 0.000 | 016 (0.9%) | 100 (1.2%) | -0.029 |
| Rheumatic Conditions | (, | - ( | | | - ( | | , | , | |
| Rheumatoid arthritis and other inflammatory polyarthropathies; n | F (4 40() | 20 (2 00() | 0.040 | 22 (4 70/) | 05 (4.40() | 0.005 | 000 (4.70() | 445 (4.20() | 0.000 |
| (%) | 5 (1.4%) | 29 (2.8%) | -0.010 | 23 (1.7%) | 86 (1.1%) | 0.005 | 028 (1.7%) | 115 (1.3%) | 0.033 |
| Osteoarthrosis; n (%) | 51 (14.0%) | 122 (11.6%) | 0.007 | 148 (11.2%) | 571 (7.6%) | 0.012 | 199 (11.8%) | 693 (8.1%) | 0.124 |
| Other rheumatic disorders (including gout); n (%) | 103 (28.4%) | 278 (26.5%) | 0.004 | 368 (27.8%) | 1,529 (20.3%) | 0.015 | 471 (27.9%) | 1,807 (21.0%) | 0.161 |
| Gout and other crystal arthropathies; n (%) | 9 (2.5%) | 21 (2.0%) | 0.003 | 20 (1.5%) | 76 (1.0%) | 0.004 | 029 (1.7%) | 097 (1.1%) | 0.051 |
| Other rheumatic disorders; n (%) | 95 (26.2%) | 263 (25.0%) | 0.002 | 353 (26.6%) | 1,473 (19.5%) | 0.015 | 448 (26.5%) | 1,736 (20.2%) | 0.149 |
| Neuro Conditions | | | | | | | | | |
| Alzheimer and other Dementia Disease ; n (%) | 5 (1.4%) | 12 (1.1%) | 0.003 | 15 (1.1%) | 46 (0.6%) | 0.005 | 020 (1.2%) | 058 (0.7%) | 0.052 |
| Seizure disorders (epilepsy); n (%) | 1 (0.3%) | 8 (0.8%) | -0.007 | 10 (0.8%) | 29 (0.4%) | 0.005 | 011 (0.7%) | 037 (0.4%) | 0.041 |
| Delirium/Psychosis; n (%) | 4 (1.1%) | 14 (1.3%) | -0.002 | 16 (1.2%) | 50 (0.7%) | 0.005 | 020 (1.2%) | 064 (0.7%) | 0.052 |
| Other Conditions | | | | | | | | | |
| Hypothyroidism; n (%) | 31 (8.5%) | 128 (12.2%) | -0.012 | 135 (10.2%) | 722 (9.6%) | 0.002 | 166 (9.8%) | 850 (9.9%) | -0.003 |
| Chronic kidney disease stages I-III; n (%) | 14 (3.9%) | 39 (3.7%) | 0.001 | 32 (2.4%) | 118 (1.6%) | 0.006 | 046 (2.7%) | 157 (1.8%) | 0.061 |
| Chronic kidney disease stages IV-V, ESRD; n (%) | 4 (1.1%) | 11 (1.0%) | 0.001 | 17 (1.3%) | 51 (0.7%) | 0.006 | 021 (1.2%) | 062 (0.7%) | 0.052 |
| COPD; n (%) | 83 (22.9%) | 152 (14.5%) | 0.019 | 294 (22.2%) | 607 (8.0%) | 0.037 | 377 (22.3%) | 759 (8.8%) | 0.379 |
| Obstructive sleep apnea; n (%) | 46 (12.7%) | 111 (10.6%) | 0.006 | 166 (12.5%) | 600 (7.9%) | 0.014 | 212 (12.6%) | 711 (8.3%) | 0.141 |
| Syncope; n (%) | 4 (1.1%) | 23 (2.2%) | -0.009 | 23 (1.7%) | 91 (1.2%) | 0.004 | 027 (1.6%) | 114 (1.3%) | 0.025 |
| Falls; n (%) | 6 (1.7%) | 21 (2.0%) | -0.002 | 6 (0.5%) | 53 (0.7%) | -0.003 | 012 (0.7%) | 074 (0.9%) | -0.022 |
| VTE; n (%) | 6 (1.7%) | 14 (1.3%) | 0.003 | 20 (1.5%) | 67 (0.9%) | 0.005 | 026 (1.5%) | 081 (0.9%) | 0.055 |
| Combined comorbidity score, 365 daysmean (sd) | 1.48 (1.68) | 1.55 (1.65) | -0.042 | 1.49 (1.58) | 1.24 (1.16) | 0.180 | 1.49 (1.60) | 1.28 (1.23) | 0.147 |
| median [IQR] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 0.000 | 1.00 [1.00, 2.00] | 1.00 [1.00, 1.00] | 0.000 | 1.49 (1.60) | 1.00 (1.23) | 0.147 |
| Frailty Score: Empirical Version 365 days as Categories | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 0.000 | 1.00 [1.00, 2.00] | 1.00 [1.00, 1.00] | 0.000 | 1.00 (1.00) | 1.00 (1.23) | 0.000 |
| <0.1 non frail; n (%) | 163 (44.9%) | 622 (59.2%) | -0.020 | 512 (38.6%) | 4,595 (60.9%) | -0.032 | 675 (40.0%) | 5,217 (60.7%) | -0.423 |
| 0.1 -< 0.2 prefrail; n (%) | 98 (27.0%) | 247 (23.5%) | 0.020 | 371 (28.0%) | 1,742 (23.1%) | 0.032 | 469 (27.8%) | 1,989 (23.1%) | 0.423 |
| > 0.2 frail; n (%) | 102 (28.1%) | 182 (17.3%) | 0.023 | 442 (33.4%) | 1,212 (16.1%) | 0.035 | 544 (32.2%) | 1,394 (16.2%) | 0.380 |
| Medication Use | 102 (20:170) | 102 (17.070) | 0.025 | (55. 170) | 1,212 (10.170) | 0.055 | 5 (52.270) | 1,00 (10.270) | 0.500 |
| Use of oral corticosteroids; n (%) | 181 (49.9%) | 507 (48.2%) | 0.002 | 663 (50.0%) | 3,950 (52.3%) | -0.003 | 844 (50.0%) | 4,457 (51.8%) | -0.036 |
| Use of antidepressants; n (%) | 95 (26.2%) | 279 (26.5%) | -0.001 | 304 (22.9%) | 1,802 (23.9%) | -0.002 | 399 (23.6%) | 2,081 (24.2%) | -0.014 |
| Use of anticonvulsants; n (%) | 27 (7.4%) | 123 (11.7%) | -0.014 | 157 (11.8%) | 649 (8.6%) | 0.010 | 184 (10.9%) | 772 (9.0%) | 0.064 |
| Use of beta blocker OR calcium channel blocker; n (%) | 72 (19.8%) | 185 (17.6%) | 0.005 | 285 (21.5%) | 964 (12.8%) | 0.021 | 357 (21.1%) | 1,149 (13.4%) | 0.205 |
| Use of PPIs; n (%) | 84 (23.1%) | 221 (21.0%) | 0.004 | 384 (29.0%) | 1,884 (25.0%) | 0.008 | 468 (27.7%) | 2,105 (24.5%) | 0.073 |
| Use of opioids; n (%) | 88 (24.2%) | 249 (23.7%) | 0.001 | 369 (27.8%) | 1,516 (20.1%) | 0.016 | 457 (27.1%) | 1,765 (20.5%) | 0.155 |
| Use of antipsychotics; n (%) | 4 (1.1%) | 27 (2.6%) | -0.011 | 28 (2.1%) | 141 (1.9%) | 0.001 | 032 (1.9%) | 168 (2.0%) | -0.007 |
| Use of anxiolytics/hypnotics; n (%) | 36 (9.9%) | 93 (8.8%) | 0.004 | 136 (10.3%) | 576 (7.6%) | 0.009 | 172 (10.2%) | 669 (7.8%) | 0.084 |
| Use of dementia meds; n (%) | 2 (0.6%) | 2 (0.2%) | 0.006 | 13 (1.0%) | 28 (0.4%) | 0.007 | 015 (0.9%) | 030 (0.3%) | 0.078 |
| Use of antiparkinsonian meds; n (%) | 4 (1.1%) | 26 (2.5%) | -0.010 | 37 (2.8%) | 107 (1.4%) | 0.010 | 041 (2.4%) | 133 (1.5%) | 0.065 |
| Use of Benzodiazepine; n (%) | 36 (9.9%) | 147 (14.0%) | -0.012 | 193 (14.6%) | 909 (12.0%) | 0.007 | 229 (13.6%) | 1,056 (12.3%) | 0.039 |
| All antidiabetic medications; n (%) | 39 (10.7%) | 117 (11.1%) | -0.001 | 176 (13.3%) | 626 (8.3%) | 0.015 | 215 (12.7%) | 743 (8.6%) | 0.133 |
| ACEI/ARB; n (%) | 112 (30.9%) | 299 (28.4%) | 0.005 | 428 (32.3%) | 1,681 (22.3%) | 0.019 | 540 (32.0%) | 1,980 (23.0%) | 0.203 |
| Use of Anticoagulants; n (%) | 12 (3.3%) | 37 (3.5%) | -0.001 | 58 (4.4%) | 176 (2.3%) | 0.011 | 070 (4.1%) | 213 (2.5%) | 0.090 |
| Use of Amiodarone; n (%) | 1 (0.3%) | 3 (0.3%) | 0.000 | 10 (0.8%) | 15 (0.2%) | 0.008 | 011 (0.7%) | 018 (0.2%) | 0.075 |
| Digoxin; n (%) | 2 (0.6%) | 5 (0.5%) | 0.001 | 20 (1.5%) | 34 (0.5%) | 0.010 | 022 (1.3%) | 039 (0.5%) | 0.085 |
| Use of Diuretics; n (%) | 85 (23.4%) | 230 (21.9%) | 0.003 | 365 (27.5%) | 1,376 (18.2%) | 0.019 | 450 (26.7%) | 1,606 (18.7%) | 0.192 |
| Use of Aspirin; n (%) | 3 (0.8%) | 3 (0.3%) | 0.007 | 10 (0.8%) | 44 (0.6%) | 0.002 | 013 (0.8%) | 047 (0.5%) | 0.037 |
| NSAIDs (NOT including aspirin); n (%) | 38 (10.5%) | 137 (13.0%) | -0.007 | 177 (13.4%) | 999 (13.2%) | 0.001 | 215 (12.7%) | 1,136 (13.2%) | -0.015 |
| HRT (Use of estrogens, progestins, androgens); n (%) | 31 (8.5%) | 140 (13.3%) | -0.015 | 160 (12.1%) | 1,209 (16.0%) | -0.010 | 191 (11.3%) | 1,349 (15.7%) | -0.129 |
| Use of Statins; n (%) | 109 (30.0%) | 287 (27.3%) | 0.005 | 428 (32.3%) | 1,626 (21.5%) | 0.021 | 537 (31.8%) | 1,913 (22.2%) | 0.218 |

| Healthcare Utilization Measures | I | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Use of any drugs claims | | | | | | | | | |
| mean (sd) | 28.06 (20.25) | 30.77 (23.08) | -0.125 | 29.03 (20.42) | 27.03 (18.93) | 0.102 | 28.82 (20.38) | 27.49 (19.48) | 0.067 |
| median [IQR] | 23.00 [13.00, 41.00] | 24.00 [16.00, 40.00] | -0.046 | 25.00 [15.00, 39.00] | 22.00 [13.00, 36.00] | 0.152 | 24.57 (20.38) | 22.24 (19.48) | 0.117 |
| Number of office visits | | | | | ,, | | . ( , | ( / | |
| mean (sd) | 11.96 (10.10) | 13.13 (11.32) | -0.109 | 12.13 (9.25) | 11.25 (10.06) | 0.091 | 12.09 (9.44) | 11.48 (10.22) | 0.062 |
| median [IQR] | 9.00 [5.00, 15.00] | 10.00 [6.00, 17.00] | -0.093 | 10.00 [5.50, 16.00] | 9.00 [5.00, 15.00] | 0.103 | 9.78 (9.44) | 9.12 (10.22) | 0.067 |
| Number of ED visits | | | | | | | , | . , | |
| mean (sd) | 0.52 (1.06) | 0.57 (1.62) | -0.037 | 0.58 (1.40) | 0.43 (1.03) | 0.122 | 0.57 (1.33) | 0.45 (1.12) | 0.098 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.000 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.000 | 0.00 (1.33) | 0.00 (1.12) | 0.000 |
| Number of hospitalizations | | | | | | | | | |
| mean (sd) | 0.12 (0.63) | 0.09 (0.41) | 0.056 | 0.54 (2.44) | 0.22 (1.55) | 0.157 | 0.45 (2.18) | 0.20 (1.46) | 0.135 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.000 | 0.00 (2.18) | 0.00 (1.46) | 0.000 |
| Recent hospitalization (-30 days to Index Rx date); n (%) | 2 (0.6%) | 16 (1.5%) | -0.009 | 29 (2.2%) | 54 (0.7%) | 0.012 | 031 (1.8%) | 070 (0.8%) | 0.088 |
| Old hospitalizations (-365 to -31 days); n (%) | 42 (11.6%) | 113 (10.8%) | 0.002 | 180 (13.6%) | 523 (6.9%) | 0.021 | 222 (13.2%) | 636 (7.4%) | 0.192 |
| Number of Pulmonologist/Allergist visits | | | | | | | | | |
| mean (sd) | 0.11 (0.59) | 0.07 (0.49) | 0.074 | 1.38 (3.13) | 2.03 (4.35) | -0.172 | 1.11 (2.79) | 1.79 (4.08) | -0.195 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.000 | 0.00 [0.00, 1.00] | 0.00 [0.00, 2.00] | 0.000 | 0.00 (2.79) | 0.00 (4.08) | 0.000 |
| Pulmonologist /allergist on CED; n (%) | 4 (1.1%) | 5 (0.5%) | 0.007 | 147 (11.1%) | 1,099 (14.6%) | -0.010 | 151 (8.9%) | 1,104 (12.8%) | -0.126 |
| Number of hospital days | | | | | | | | | |
| mean (sd) | 1.51 (10.26) | 0.74 (4.89) | 0.096 | 0.54 (2.44) | 0.22 (1.55) | 0.157 | 0.75 (5.22) | 0.28 (2.24) | 0.117 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.000 | 0.00 (5.22) | 0.00 (2.24) | 0.000 |
| Occurrence of basic or comprehensive metabolic blood chemistry | 149 (41.0%) | 406 (38.6%) | 0.004 | 434 (32.8%) | 2,074 (27.5%) | 0.010 | 583 (34.5%) | 2,480 (28.8%) | 0.123 |
| test; n (%) | 149 (41.0%) | 400 (38.0%) | 0.004 | 434 (32.6%) | 2,074 (27.3%) | 0.010 | 363 (34.3%) | 2,460 (26.6%) | 0.123 |
| Number of HbA1C test ordered | | | | | | | | | |
| mean (sd) | 0.51 (1.00) | 0.55 (1.12) | -0.038 | 0.45 (1.00) | 0.38 (0.91) | 0.073 | 0.46 (1.00) | 0.40 (0.94) | 0.062 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.000 | 0.00 (1.00) | 0.00 (0.94) | 0.000 |
| Flexible Sigmoidoscopy or colonoscopy or CT virtual colonoscopy; n (%) | 18 (5.0%) | 34 (3.2%) | 0.009 | 70 (5.3%) | 291 (3.9%) | 0.007 | 088 (5.2%) | 325 (3.8%) | 0.068 |
| Number of Mammograms (Breast cancer screening); n (%) | 46 (12.7%) | 151 (14.4%) | -0.005 | 175 (13.2%) | 1,091 (14.5%) | -0.003 | 221 (13.1%) | 1,242 (14.4%) | -0.038 |
| Number of Pap smear (Cervical cancer screening); n (%) | 29 (8.0%) | 110 (10.5%) | -0.008 | 107 (8.1%) | 814 (10.8%) | -0.009 | 136 (8.1%) | 924 (10.7%) | -0.089 |
| Flu vaccine; n (%) | 66 (18.2%) | 212 (20.2%) | -0.005 | 193 (14.6%) | 1,316 (17.4%) | -0.007 | 259 (15.3%) | 1,528 (17.8%) | -0.067 |
| Pneumococcal vaccine; n (%) | 10 (2.8%) | 96 (9.1%) | -0.026 | 42 (3.2%) | 622 (8.2%) | -0.021 | 052 (3.1%) | 718 (8.3%) | -0.226 |
| Copay for pharmacy cost (charges in U.S. \$) | , , | , , | | , , | | | | | |
| mean (sd) | 38.10 (33.36) | 37.67 (31.88) | 0.013 | 34.89 (33.21) | 26.35 (23.40) | 0.297 | 35.58 (33.24) | 27.73 (24.59) | 0.268 |
| median [IQR] | 30.00 [18.95, 47.48] | 31.94 [17.50, 50.14] | -0.059 | 28.41 [15.61, 43.95] | 22.44 [11.87, 35.15] | 0.208 | 28.75 (33.24) | 23.60 (24.59) | 0.176 |
| Business Type | | | | | | | | | |
| Commercial; n (%) | 312 (86.0%) | 835 (79.4%) | 0.007 | NA | NA | NA | NA | NA | NA |
| Medicare; n (%) | 51 (14.0%) | 216 (20.6%) | -0.016 | NA | NA | NA | NA | NA | NA |
| Insurance Plan Type | | | | | | | | | |
| Comprehensive; n (%) | NA | NA | NA | 188 (14.2%) | 494 (6.5%) | 0.024 | NA | NA | NA |
| HMO; n (%) | NA | NA | NA | 150 (11.3%) | 1,357 (18.0%) | -0.018 | NA | NA | NA |
| PPO; n (%) | NA | NA | NA | 758 (57.2%) | 4,103 (54.4%) | 0.004 | NA | NA | NA |
| Others; n (%) | NA | NA | NA | 229 (17.3%) | 1,595 (21.1%) | -0.009 | NA | NA | NA |
| SABA; n (%) | 164 (45.2%) | 615 (58.5%) | -0.019 | 773 (58.3%) | 4,829 (64.0%) | -0.007 | 937 (55.5%) | 5,444 (63.3%) | -0.159 |
| SAMA; n (%) | 16 (4.4%) | 33 (3.1%) | 0.007 | 60 (4.5%) | 254 (3.4%) | 0.006 | 076 (4.5%) | 287 (3.3%) | 0.062 |
| SABA/SAMA; n (%) | 25 (6.9%) | 45 (4.3%) | 0.011 | 118 (8.9%) | 263 (3.5%) | 0.022 | 143 (8.5%) | 308 (3.6%) | 0.207 |
| ICS; n (%) | 332 (91.5%) | 442 (42.1%) | 0.061 | 1,211 (91.4%) | 4,052 (53.7%) | 0.044 | 1,543 (91.4%) | 4,494 (52.3%) | 0.965 |
| LABA without formoterol; n (%) | 21 (5.8%) | 3 (0.3%) | 0.032 | 73 (5.5%) | 57 (0.8%) | 0.026 | 094 (5.6%) | 060 (0.7%) | 0.283 |
| LAMA; n (%) | 46 (12.7%) | 70 (6.7%) | 0.019 | 187 (14.1%) | 378 (5.0%) | 0.029 | 233 (13.8%) | 448 (5.2%) | 0.297 |
| LABA/ICS without mometasone-formoterol; n (%) | 91 (25.1%) | 430 (40.9%) | -0.028 | 326 (24.6%) | 3,189 (42.2%) | -0.031 | 417 (24.7%) | 3,619 (42.1%) | -0.375 |
| Blood eosinophilia test ; n (%) | 0 (0.0%) | 5 (0.5%) | -0.010 | 4 (0.3%) | 15 (0.2%) | 0.002 | 004 (0.2%) | 020 (0.2%) | 0.000 |
| Serum immunoglobulin E (IgE) level test; n (%) | 7 (1.9%) | 28 (2.7%) | -0.005 | 29 (2.2%) | 293 (3.9%) | -0.010 | 036 (2.1%) | 321 (3.7%) | -0.095 |
| H2 blocker; n (%) | 5 (1.4%) | 27 (2.6%) | -0.008 | 44 (3.3%) | 311 (4.1%) | -0.004 | 049 (2.9%) | 338 (3.9%) | -0.055 |
| Oxygen codes; n (%) | 11 (3.0%) | 15 (1.4%) | 0.011 | 40 (3.0%) | 46 (0.6%) | 0.018 | 051 (3.0%) | 061 (0.7%) | 0.171 |
| Respiratory arrest/dependence on oxygen; n (%) | 8 (2.2%) | 6 (0.6%) | 0.014 | 10 (0.8%) | 25 (0.3%) | 0.007 | 018 (1.1%) | 031 (0.4%) | 0.081 |

Aetion link to Optum results: https://bwh-dope.aetion.com/projects/details/1659/rwrs/68458
Aetion link to Marketscan results: https://bwh-dope.aetion.com/projects/details/1658/rwrs/68457

| | | | PS-match | ned | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Optum | | - C .Hatel | | ketscan | | POOLED | | |
| Variable | Formoterol fumarate<br>10 mcg | Mometasone<br>furoate/formoterol<br>fumarate | St. Diff. | Formoterol fumarate<br>10 mcg | Mometasone<br>furoate/formoterol<br>fumarate | St. Diff. | Formoterol fumarate<br>10 mcg | Mometasone<br>furoate/formoterol<br>fumarate | St. Diff. |
| Number of patients | 165 | 165 | 5 | 919 | 919 | | 1,084 | 1,08 | ţ |
| Year of Cohort Entry Date | | | | | | | | | |
| 2010; n (%) | 11 (6.7%) | 7 (4.2%) | 0.0107 | 73 (7.9%) | 89 (9.7%) | -0.0061 | 084 (7.7%) | 096 (8.9%) | -0.044 |
| 2011; n (%) | 33 (20.0%) | 41 (24.8%) | -0.0102 | 276 (30.0%) | 247 (26.9%) | 0.0058 | 309 (28.5%) | 288 (26.6%) | 0.043 |
| 2012; n (%) | 40 (24.2%) | 43 (26.1%) | -0.0038 | 210 (22.9%) | 223 (24.3%) | -0.0029 | 250 (23.1%) | 266 (24.5%) | -0.033 |
| 2013; n (%) | 34 (20.6%) | 25 (15.2%) | 0.0128 | 131 (14.3%) | 136 (14.8%) | -0.0013 | 165 (15.2%) | 161 (14.9%) | 0.008 |
| 2014; n (%) | 28 (17.0%) | 26 (15.8%) | 0.0030 | 140 (15.2%) | 131 (14.3%) | 0.0023 | 168 (15.5%) | 157 (14.5%) | 0.028 |
| 2015; n (%) | 15 (9.1%) | 16 (9.7%) | -0.0020 | 76 (8.3%) | 78 (8.5%) | -0.0007 | 091 (8.4%) | 094 (8.7%) | -0.011 |
| 2016; n (%) | 4 (2.4%) | 7 (4.2%) | -0.0099 | 13 (1.4%) | 15 (1.6%) | -0.0016 | 017 (1.6%) | 022 (2.0%) | -0.030 |
| 2017; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 000 (0.0%) | 000 (0.0%) | #DIV/0! |
| 2018; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 000 (0.0%) | 000 (0.0%) | #DIV/0! |
| 2019; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | NA | NA | NA | NA | NA , | NA |
| 2020; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | NA | NA | NA | NA | NA | NA |
| Age* | , , | , , | • | | | | | | |
| mean (sd) | 52.62 (15.47) | 53.08 (16.38) | -0.0289 | 53.73 (15.97) | 53.63 (17.30) | 0.0060 | 53.56 (15.90) | 53.55 (17.16) | 0.001 |
| median [IQR] | 54.00 [45.00, 63.50] | 54.00 [44.00, 63.50] | 0.0000 | 57.00 [45.00, 63.00] | 56.00 [44.00, 64.00] | 0.0601 | 56.54 (15.90) | 55.70 (17.16) | 0.051 |
| Age categories | | | | | | | (, | | |
| 12-17; n (%) | 4 (2.4%) | 7 (4.2%) | -0.0099 | 32 (3.5%) | 52 (5.7%) | -0.0103 | 036 (3.3%) | 059 (5.4%) | -0.103 |
| 18-39; n (%) | 27 (16.4%) | 23 (13.9%) | 0.0064 | 114 (12.4%) | 120 (13.1%) | -0.0020 | 141 (13.0%) | 143 (13.2%) | -0.006 |
| 40 - 64; n (%) | 95 (57.6%) | 100 (60.6%) | -0.0039 | 580 (63.1%) | 540 (58.8%) | 0.0055 | 675 (62.3%) | 640 (59.0%) | 0.068 |
| >= 65; n (%) | 39 (23.6%) | 35 (21.2%) | 0.0051 | 193 (21.0%) | 207 (22.5%) | -0.0032 | 232 (21.4%) | 242 (22.3%) | -0.022 |
| Geographic Region* | 39 (23.0%) | 33 (21.270) | 0.0031 | 133 (21.070) | 207 (22.570) | -0.0032 | 232 (21.470) | 242 (22.370) | -0.022 |
| Northeast; n (%) | 22 (13.3%) | 19 (11.5%) | 0.0051 | 225 (24.5%) | 227 (24.7%) | -0.0004 | 247 (22.8%) | 246 (22.7%) | 0.002 |
| | 68 (41.2%) | 71 (43.0%) | -0.0028 | 293 (31.9%) | 294 (32.0%) | -0.0004 | 361 (33.3%) | 365 (33.7%) | -0.002 |
| South; n (%) | | | | | | 0.0002 | | | 0.019 |
| Midwest; n (%) | 44 (26.7%)<br>31 (18.8%) | 42 (25.5%)<br>33 (20.0%) | 0.0024<br>-0.0027 | 213 (23.2%)<br>172 (18.7%) | 206 (22.4%)<br>176 (19.2%) | -0.0017 | 257 (23.7%)<br>203 (18.7%) | 248 (22.9%)<br>209 (19.3%) | -0.019 |
| West; n (%) | | 33 (20.0%)<br>NA | | | | 0.0001 | | | |
| Unknown/Missing; n (%) | NA | NA | NA | 16 (1.7%) | 16 (1.7%) | 0.0000 | NA | NA | NA |
| Metropolitan Statistical Area* | N.O. | N/A | | 742 (00 70/) | 762 (02 00/) | 0.0000 | N/A | N1.0 | |
| Urban; n (%) | NA<br>NA | NA<br>NA | NA | 742 (80.7%) | 763 (83.0%) | -0.0026 | NA | NA | NA |
| Rural; n (%) | NA<br>NA | NA<br>NA | NA | 2 (0.2%) | 5 (0.5%) | -0.0051 | NA | NA | NA |
| Unknown/Missing; n (%) | NA | NA | NA | 175 (19.0%) | 151 (16.4%) | 0.0062 | NA | NA | NA |
| General Health Related Measures | - (() | | | * ** *** | | | | | |
| Alcohol/Drug abuse or dependence ; n (%) | 3 (1.8%) | 2 (1.2%) | 0.0049 | 9 (1.0%) | 12 (1.3%) | -0.0028 | 012 (1.1%) | 014 (1.3%) | -0.018 |
| Obesity or Overweight; n (%)* | 15 (9.1%) | 20 (12.1%) | -0.0092 | 77 (8.4%) | 87 (9.5%) | -0.0037 | 092 (8.5%) | 107 (9.9%) | -0.048 |
| Obesity; n (%) | 13 (7.9%) | 17 (10.3%) | -0.0080 | 68 (7.4%) | 77 (8.4%) | -0.0036 | 081 (7.5%) | 094 (8.7%) | -0.044 |
| Overweight; n (%) | 2 (1.2%) | 3 (1.8%) | -0.0049 | 12 (1.3%) | 10 (1.1%) | 0.0018 | 014 (1.3%) | 013 (1.2%) | 0.009 |
| Cardiovascular Measures | | | | | | | | | |
| Hypertension; n (%)* | 63 (38.2%) | 60 (36.4%) | 0.0030 | 325 (35.4%) | 332 (36.1%) | -0.0012 | 388 (35.8%) | 392 (36.2%) | -0.008 |
| Hyperlipidemia; n (%)* | 54 (32.7%) | 49 (29.7%) | 0.0054 | 254 (27.6%) | 273 (29.7%) | -0.0039 | 308 (28.4%) | 322 (29.7%) | -0.029 |
| MI, angina, Coronary atherosclerosis and other forms of chronic | 12 (7.3%) | 9 (5.5%) | 0.0071 | 75 (8.2%) | 83 (9.0%) | -0.0027 | 087 (8.0%) | 092 (8.5%) | -0.018 |
| ischemic heart disease; n (%)* | | | | | | | | | |
| Old MI; n (%) | 2 (1.2%) | 1 (0.6%) | 0.0063 | 5 (0.5%) | 4 (0.4%) | 0.0015 | 007 (0.6%) | 005 (0.5%) | 0.014 |
| Acute MI; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 2 (0.2%) | 2 (0.2%) | 0.0000 | 002 (0.2%) | 002 (0.2%) | 0.000 |
| Stable angina; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 10 (1.1%) | 7 (0.8%) | 0.0031 | 010 (0.9%) | 007 (0.6%) | 0.035 |
| Coronary atherosclerosis and other forms of chronic ischemic heart disease; n (%) | 12 (7.3%) | 9 (5.5%) | 0.0071 | 68 (7.4%) | 72 (7.8%) | -0.0015 | 080 (7.4%) | 081 (7.5%) | -0.004 |
| History of CABG or PTCA; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 7 (0.8%) | 5 (0.5%) | 0.0037 | 007 (0.6%) | 005 (0.5%) | 0.014 |
| Cerebrovascular disease (Stroke, TIA, Late effects); n (%)* | 2 (1.2%) | 3 (1.8%) | -0.0049 | 12 (1.3%) | 9 (1.0%) | 0.0028 | 014 (1.3%) | 012 (1.1%) | 0.018 |
| Stroke (Ischemic or hemorrhagic); n (%) | 2 (1.2%) | 0 (0.0%) | 0.0155 | 7 (0.8%) | 6 (0.7%) | 0.0012 | 009 (0.8%) | 006 (0.6%) | 0.024 |
| TIA; n (%) | 0 (0.0%) | 2 (1.2%) | -0.0155 | 6 (0.7%) | 3 (0.3%) | 0.0057 | 006 (0.6%) | 005 (0.5%) | 0.014 |
| Late effects of cerebrovascular disease; n (%) | 0 (0.0%) | 1 (0.6%) | -0.0110 | 5 (0.5%) | 1 (0.1%) | 0.0073 | 005 (0.5%) | 002 (0.2%) | 0.051 |
| Atrial fibrillation and Other cardiac dysrhythmia; n (%)* | 10 (6.1%) | 12 (7.3%) | -0.0046 | 64 (7.0%) | 62 (6.7%) | 0.0011 | 074 (6.8%) | 074 (6.8%) | 0.000 |
| Atrial fibrillation; n (%) | 3 (1.8%) | 6 (3.6%) | -0.0110 | 38 (4.1%) | 32 (3.5%) | 0.0031 | 041 (3.8%) | 038 (3.5%) | 0.016 |
| Other cardiac dysrhythmia; n (%) | 7 (4.2%) | 8 (4.8%) | -0.0028 | 39 (4.2%) | 39 (4.2%) | 0.0000 | 046 (4.2%) | 047 (4.3%) | -0.005 |
| Diabetes Related Measures | | | | | | | | | |
| Diabetes with or w/o complications; n (%)* | 23 (13.9%) | 25 (15.2%) | -0.0034 | 130 (14.1%) | 126 (13.7%) | 0.0011 | 153 (14.1%) | 151 (13.9%) | 0.006 |
| | • | | | • • | • • | | | | |

| | • | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Diabetes mellitus without mention of complications; n (%) | 23 (13.9%) | 25 (15.2%) | -0.0034 | 124 (13.5%) | 119 (12.9%) | 0.0017 | 147 (13.6%) | 144 (13.3%) | 0.009 |
| Diabetes with specified complications; n (%) | 4 (2.4%) | 7 (4.2%) | -0.0099 | 29 (3.2%) | 20 (2.2%) | 0.0061 | 033 (3.0%) | 027 (2.5%) | 0.031 |
| Diabetes with unspecified complications; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 5 (0.5%) | 3 (0.3%) | 0.0032 | 005 (0.5%) | 003 (0.3%) | 0.032 |
| GI Conditions | / // | / // | | | | | | | |
| GERD; n (%)* | 22 (13.3%) | 28 (17.0%) | -0.0095 | 120 (13.1%) | 123 (13.4%) | -0.0008 | 142 (13.1%) | 151 (13.9%) | -0.023 |
| Upper GI (Diseases of esophagus, stomach and duodenum including GERD); n (%) | 25 (15.2%) | 31 (18.8%) | -0.0087 | 152 (16.5%) | 161 (17.5%) | -0.0024 | 177 (16.3%) | 192 (17.7%) | -0.037 |
| GI bleeding; n (%)* | 3 (1.8%) | 2 (1.2%) | 0.0049 | 14 (1.5%) | 12 (1.3%) | 0.0017 | 017 (1.6%) | 014 (1.3%) | 0.025 |
| Non-infective enteritis and colitis; n (%) | 6 (3.6%) | 10 (6.1%) | -0.0114 | 40 (4.4%) | 37 (4.0%) | 0.0020 | 046 (4.2%) | 047 (4.3%) | -0.005 |
| Intraoperative and postprocedural complications and disorders of | 2 (1.2%) | 2 (1.2%) | 0.0000 | 16 (1.7%) | 17 (1.8%) | -0.0008 | 018 (1.7%) | 019 (1.8%) | -0.008 |
| digestive system; n (%) | | | | | | | | | |
| Disorders of gallbladder, biliary tract and pancreas; n (%)* | 1 (0.6%) | 0 (0.0%) | 0.0110 | 11 (1.2%) | 7 (0.8%) | 0.0040 | 012 (1.1%) | 007 (0.6%) | 0.054 |
| Rheumatic Conditions Rheumatoid arthritis and other inflammatory polyarthropathies; n | | | | | | | | | |
| (%)* | 2 (1.2%) | 3 (1.8%) | -0.0049 | 17 (1.8%) | 14 (1.5%) | 0.0023 | 019 (1.8%) | 017 (1.6%) | 0.015 |
| Osteoarthrosis; n (%)* | 21 (12.7%) | 22 (13.3%) | -0.0017 | 90 (9.8%) | 91 (9.9%) | -0.0003 | 111 (10.2%) | 113 (10.4%) | -0.007 |
| Other rheumatic disorders (including gout); n (%)* | 40 (24.2%) | 46 (27.9%) | -0.0073 | 234 (25.5%) | 249 (27.1%) | -0.0031 | 274 (25.3%) | 295 (27.2%) | -0.043 |
| Gout and other crystal arthropathies; n (%) | 2 (1.2%) | 4 (2.4%) | -0.0089 | 14 (1.5%) | 20 (2.2%) | -0.0051 | 016 (1.5%) | 024 (2.2%) | -0.052 |
| Other rheumatic disorders; n (%) | 38 (23.0%) | 43 (26.1%) | -0.0063 | 225 (24.5%) | 233 (25.4%) | -0.0018 | 263 (24.3%) | 276 (25.5%) | -0.028 |
| Neuro Conditions* | | | | | | | | | |
| Alzheimer and other Dementia Disease ; n (%) | 1 (0.6%) | 2 (1.2%) | -0.0063 | 7 (0.8%) | 11 (1.2%) | -0.0040 | 008 (0.7%) | 013 (1.2%) | -0.052 |
| Seizure disorders (epilepsy); n (%) | 0 (0.0%) | 1 (0.6%) | -0.0110 | 6 (0.7%) | 8 (0.9%) | -0.0022 | 006 (0.6%) | 009 (0.8%) | -0.024 |
| Delirium/Psychosis; n (%) | 1 (0.6%) | 1 (0.6%) | 0.0000 | 8 (0.9%) | 9 (1.0%) | -0.0010 | 009 (0.8%) | 010 (0.9%) | -0.011 |
| Other Conditions | | | | | | | | | |
| Hypothyroidism; n (%)* | 12 (7.3%) | 13 (7.9%) | -0.0022 | 99 (10.8%) | 110 (12.0%) | -0.0036 | 111 (10.2%) | 123 (11.3%) | -0.036 |
| Chronic kidney disease stages I-III; n (%)* | 4 (2.4%) | 4 (2.4%) | 0.0000 | 15 (1.6%) | 19 (2.1%) | -0.0037 | 019 (1.8%) | 023 (2.1%) | -0.022 |
| Chronic kidney disease stages IV-V, ESRD; n (%) | 1 (0.6%) | 2 (1.2%) | -0.0063 | 7 (0.8%) | 10 (1.1%) | -0.0031 | 008 (0.7%) | 012 (1.1%) | -0.042 |
| COPD; n (%)* | 25 (15.2%) | 29 (17.6%) | -0.0059 | 147 (16.0%) | 160 (17.4%) | -0.0034 | 172 (15.9%) | 189 (17.4%) | -0.040 |
| Obstructive sleep apnea; n (%)* | 15 (9.1%) | 17 (10.3%) | -0.0039 | 108 (11.8%) | 117 (12.7%) | -0.0026 | 123 (11.3%) | 134 (12.4%) | -0.034 |
| Syncope; n (%) | 3 (1.8%) | 2 (1.2%) | 0.0049 | 12 (1.3%) | 16 (1.7%) | -0.0033 | 015 (1.4%) | 018 (1.7%) | -0.024 |
| Falls; n (%)<br>VTE; n (%)* | 1 (0.6%) | 4 (2.4%) | -0.0147<br>-0.0041 | 5 (0.5%) | 3 (0.3%) | 0.0032<br>0.0045 | 006 (0.6%)<br>017 (1.6%) | 007 (0.6%) | 0.000<br>0.034 |
| Combined comorbidity score, 365 days* | 3 (1.8%) | 4 (2.4%) | -0.0041 | 14 (1.5%) | 9 (1.0%) | 0.0045 | 017 (1.6%) | 013 (1.2%) | 0.034 |
| mean (sd) | 1.26 (1.30) | 1.34 (1.15) | -0.0652 | 1.38 (1.39) | 1.42 (1.52) | -0.0275 | 1.36 (1.38) | 1.41 (1.47) | -0.035 |
| median [IQR] | 1.00 [1.00, 1.00] | 1.00 [1.00, 2.00] | 0.0000 | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 0.0000 | 1.00 (1.38) | 1.00 (1.47) | 0.000 |
| Frailty Score: Empirical Version 365 days as Categories* | 1.00 (1.00) 1.00) | 1.00 (1.00) 2.00) | 0.0000 | 1.00 (1.00, 2.00) | 1.00 (1.00, 1.00) | 0.0000 | 1.00 (1.50) | 1.00 (1.17) | 0.000 |
| <0.1 non frail; n (%) | 81 (49.1%) | 90 (54.5%) | -0.0075 | 409 (44.5%) | 406 (44.2%) | 0.0005 | 490 (45.2%) | 496 (45.8%) | -0.012 |
| 0.1 -< 0.2 prefrail; n (%) | 45 (27.3%) | 39 (23.6%) | 0.0073 | 261 (28.4%) | 261 (28.4%) | 0.0000 | 306 (28.2%) | 300 (27.7%) | 0.011 |
| > 0.2 frail; n (%) | 39 (23.6%) | 36 (21.8%) | 0.0038 | 249 (27.1%) | 252 (27.4%) | -0.0006 | 288 (26.6%) | 288 (26.6%) | 0.000 |
| Medication Use | | | | | | | | | |
| Use of oral corticosteroids; n (%)* | 82 (49.7%) | 79 (47.9%) | 0.0026 | 458 (49.8%) | 475 (51.7%) | -0.0027 | 540 (49.8%) | 554 (51.1%) | -0.026 |
| Use of antidepressants; n (%)* | 40 (24.2%) | 36 (21.8%) | 0.0050 | 223 (24.3%) | 228 (24.8%) | -0.0010 | 263 (24.3%) | 264 (24.4%) | -0.002 |
| Use of anticonvulsants; n (%)* | 17 (10.3%) | 15 (9.1%) | 0.0039 | 101 (11.0%) | 100 (10.9%) | 0.0003 | 118 (10.9%) | 115 (10.6%) | 0.010 |
| Use of beta blocker OR calcium channel blocker; n (%)* | 24 (14.5%) | 17 (10.3%) | 0.0119 | 166 (18.1%) | 164 (17.8%) | 0.0007 | 190 (17.5%) | 181 (16.7%) | 0.021 |
| Use of PPIs; n (%)* | 37 (22.4%) | 39 (23.6%) | -0.0025 | 267 (29.1%) | 263 (28.6%) | 0.0009 | 304 (28.0%) | 302 (27.9%) | 0.002 |
| Use of opioids; n (%)* | 37 (22.4%) | 42 (25.5%) | -0.0063 | 245 (26.7%) | 235 (25.6%) | 0.0022 | 282 (26.0%) | 277 (25.6%) | 0.009 |
| Use of antipsychotics; n (%)* | 2 (1.2%) | 1 (0.6%) | 0.0063 | 16 (1.7%) | 17 (1.8%) | -0.0008 | 018 (1.7%) | 018 (1.7%) | 0.000 |
| Use of anxiolytics/hypnotics; n (%)* | 15 (9.1%) | 15 (9.1%) | 0.0000 | 84 (9.1%) | 96 (10.4%) | -0.0042 | 099 (9.1%) | 111 (10.2%) | -0.037 |
| Use of dementia meds; n (%)* | 0 (0.0%) | 1 (0.6%) | -0.0110 | 6 (0.7%) | 9 (1.0%) | -0.0033 | 006 (0.6%) | 010 (0.9%) | -0.035 |
| Use of antiparkinsonian meds; n (%)* Use of Benzodiazepine; n (%)* | 2 (1.2%) | 3 (1.8%) | -0.0049<br>-0.0041 | 23 (2.5%) | 25 (2.7%) | -0.0012<br>-0.0005 | 025 (2.3%) | 028 (2.6%) | -0.019<br>-0.012 |
| All antidiabetic medications; n (%)* | 13 (7.9%)<br>17 (10.3%) | 15 (9.1%)<br>20 (12.1%) | -0.0041 | 137 (14.9%)<br>109 (11.9%) | 139 (15.1%)<br>100 (10.9%) | 0.0003 | 150 (13.8%)<br>126 (11.6%) | 154 (14.2%)<br>120 (11.1%) | 0.012 |
| ACEI/ARB; n (%)* | 48 (29.1%) | 40 (24.2%) | 0.0034 | 269 (29.3%) | 256 (27.9%) | 0.0030 | 317 (29.2%) | 296 (27.3%) | 0.010 |
| Use of Anticoagulants; n (%)* | 3 (1.8%) | 5 (3.0%) | -0.0033 | 36 (3.9%) | 33 (3.6%) | 0.0020 | 039 (3.6%) | 038 (3.5%) | 0.042 |
| Use of Amiodarone; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 4 (0.4%) | 6 (0.7%) | -0.0040 | 004 (0.4%) | 006 (0.6%) | -0.028 |
| Digoxin; n (%) | 1 (0.6%) | 1 (0.6%) | 0.0000 | 9 (1.0%) | 10 (1.1%) | -0.0010 | 010 (0.9%) | 011 (1.0%) | -0.010 |
| Use of Diuretics; n (%)* | 38 (23.0%) | 31 (18.8%) | 0.0092 | 215 (23.4%) | 215 (23.4%) | 0.0000 | 253 (23.3%) | 246 (22.7%) | 0.014 |
| Use of Aspirin; n (%) | 1 (0.6%) | 0 (0.0%) | 0.0110 | 7 (0.8%) | 7 (0.8%) | 0.0000 | 008 (0.7%) | 007 (0.6%) | 0.012 |
| NSAIDs (NOT including aspirin); n (%) | 18 (10.9%) | 24 (14.5%) | -0.0101 | 115 (12.5%) | 145 (15.8%) | -0.0088 | 133 (12.3%) | 169 (15.6%) | -0.095 |
| HRT (Use of estrogens, progestins, androgens); n (%)* | 19 (11.5%) | 19 (11.5%) | 0.0000 | 122 (13.3%) | 128 (13.9%) | -0.0016 | 141 (13.0%) | 147 (13.6%) | -0.018 |
| Use of Statins ; n (%)* | 45 (27.3%) | 46 (27.9%) | -0.0011 | 262 (28.5%) | 280 (30.5%) | -0.0037 | 307 (28.3%) | 326 (30.1%) | -0.040 |
| | • | • | | • | | | • | | |

| In an arm of the | Ī | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Healthcare Utilization Measures | | | | | | | | | |
| Use of any drugs claims* | | | | | | | | | |
| mean (sd) | 28.42 (20.68) | 28.33 (20.78) | 0.0043 | 28.80 (20.50) | 29.10 (20.30) | -0.0147 | 28.74 (20.53) | 28.98 (20.37) | -0.012 |
| median [IQR] | 22.00 [13.00, 40.00] | 21.00 [14.00, 36.00] | 0.0482 | 24.00 [14.00, 38.00] | 25.00 [15.00, 38.00] | -0.0490 | 23.70 (20.53) | 24.39 (20.37) | -0.034 |
| Number of office visits* | | | | | | | | | |
| mean (sd) | 11.42 (9.14) | 11.35 (9.38) | 0.0076 | 12.04 (9.09) | 12.12 (9.09) | -0.0088 | 11.95 (9.10) | 12.00 (9.13) | -0.005 |
| median [IQR] | 9.00 [5.00, 15.00] | 8.00 [5.00, 13.50] | 0.1080 | 10.00 [5.00, 16.00] | 10.00 [6.00, 15.00] | 0.0000 | 9.85 (9.10) | 9.70 (9.13) | 0.016 |
| Number of ED visits* | | | | | | | | | |
| mean (sd) | 0.41 (0.86) | 0.38 (1.00) | 0.0322 | 0.52 (1.28) | 0.49 (1.20) | 0.0242 | 0.50 (1.23) | 0.47 (1.17) | 0.025 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.0000 | 0.00 (1.23) | 0.00 (1.17) | 0.000 |
| Number of hospitalizations* | | | | | | | | | |
| mean (sd) | 0.04 (0.23) | 0.05 (0.27) | -0.0399 | 0.39 (2.13) | 0.34 (1.75) | 0.0257 | 0.34 (1.96) | 0.30 (1.62) | 0.022 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (1.96) | 0.00 (1.62) | 0.000 |
| Recent hospitalization (-30 days to Index Rx date); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 11 (1.2%) | 12 (1.3%) | -0.0009 | 011 (1.0%) | 012 (1.1%) | -0.010 |
| Old hospitalizations (-365 to -31 days); n (%) | 15 (9.1%) | 11 (6.7%) | 0.0085 | 97 (10.6%) | 93 (10.1%) | 0.0016 | 112 (10.3%) | 104 (9.6%) | 0.023 |
| Number of Pulmonologist/Allergist visits* | | | | | | | | | |
| mean (sd) | 0.10 (0.45) | 0.08 (0.43) | 0.0454 | 1.61 (3.53) | 1.79 (3.40) | -0.0519 | 1.38 (3.26) | 1.53 (3.14) | -0.047 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | -0.2885 | 0.00 (3.26) | 0.85 (3.14) | -0.266 |
| Pulmonologist /allergist on CED; n (%)* | 2 (1.2%) | 2 (1.2%) | 0.0000 | 117 (12.7%) | 136 (14.8%) | -0.0057 | 119 (11.0%) | 138 (12.7%) | -0.053 |
| Number of hospital days* | | | | | | | | | |
| mean (sd) | 0.23 (1.38) | 0.45 (3.12) | -0.0912 | 0.39 (2.13) | 0.34 (1.75) | 0.0257 | 0.37 (2.03) | 0.36 (2.02) | 0.005 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (2.03) | 0.00 (2.02) | 0.000 |
| Occurrence of basic or comprehensive metabolic blood chemistry | E0 (2E 20/) | CO (2C 40/) | -0.0020 | 200 (21 69/) | 206 (21 10/) | 0.0009 | 249 (22 49/) | 246 (24.00/) | 0.004 |
| test; n (%)* | 58 (35.2%) | 60 (36.4%) | -0.0020 | 290 (31.6%) | 286 (31.1%) | 0.0009 | 348 (32.1%) | 346 (31.9%) | 0.004 |
| Number of HbA1C test ordered* | | | | | | | | | |
| mean (sd) | 0.42 (0.88) | 0.56 (1.23) | -0.1309 | 0.42 (0.95) | 0.39 (0.92) | 0.0321 | 0.42 (0.94) | 0.42 (0.97) | 0.000 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (0.94) | 0.00 (0.97) | 0.000 |
| Flexible Sigmoidoscopy or colonoscopy or CT virtual colonoscopy; | 2 (4 00/) | C (2, C0() | 0.0110 | 40 (F 20/) | F7 (C 20() | 0.0020 | 052 (4.00/) | 0.63 (5.00/) | -0.045 |
| n (%)* | 3 (1.8%) | 6 (3.6%) | -0.0110 | 49 (5.3%) | 57 (6.2%) | -0.0038 | 052 (4.8%) | 063 (5.8%) | -0.045 |
| Number of Mammograms (Breast cancer screening); n (%)* | 21 (12.7%) | 22 (13.3%) | -0.0017 | 131 (14.3%) | 142 (15.5%) | -0.0031 | 152 (14.0%) | 164 (15.1%) | -0.031 |
| Number of Pap smear (Cervical cancer screening); n (%)* | 14 (8.5%) | 14 (8.5%) | 0.0000 | 88 (9.6%) | 78 (8.5%) | 0.0037 | 102 (9.4%) | 092 (8.5%) | 0.032 |
| Flu vaccine; n (%)* | 29 (17.6%) | 27 (16.4%) | 0.0029 | 139 (15.1%) | 144 (15.7%) | -0.0015 | 168 (15.5%) | 171 (15.8%) | -0.008 |
| Pneumococcal vaccine; n (%)* | 7 (4.2%) | 8 (4.8%) | -0.0028 | 37 (4.0%) | 37 (4.0%) | 0.0000 | 044 (4.1%) | 045 (4.2%) | -0.005 |
| Copay for pharmacy cost (charges in U.S. \$)* | | | | | | | | | |
| mean (sd) | 36.76 (34.33) | 35.41 (28.84) | 0.0426 | 32.44 (29.37) | 32.24 (28.07) | 0.0070 | 33.10 (30.17) | 32.72 (28.19) | 0.013 |
| median [IQR] | 28.33 [18.09, 45.06] | 29.38 [17.97, 48.77] | -0.0331 | 27.29 [14.61, 42.08] | 27.00 [16.00, 41.79] | 0.0101 | 27.45 (30.17) | 27.36 (28.19) | 0.003 |
| Business Type* | | | | | | | | | |
| Commercial; n (%) | 140 (84.8%) | 136 (82.4%) | 0.0026 | NA | NA | NA | NA | NA | NA |
| Medicare; n (%) | 25 (15.2%) | 29 (17.6%) | -0.0059 | NA | NA | NA | NA | NA | NA |
| Insurance Plan Type* | | | | | | | | | |
| Comprehensive; n (%) | NA | NA | NA | 96 (10.4%) | 96 (10.4%) | 0.0000 | NA | NA | NA |
| HMO; n (%) | NA | NA | NA | 111 (12.1%) | 102 (11.1%) | 0.0029 | NA | NA | NA |
| PPO; n (%) | NA | NA | NA | 543 (59.1%) | 551 (60.0%) | -0.0012 | NA | NA | NA |
| Others; n (%) | NA | NA | NA | 169 (18.4%) | 170 (18.5%) | -0.0002 | NA | NA | NA |
| SABA; n (%)* | 87 (52.7%) | 86 (52.1%) | 0.0008 | 555 (60.4%) | 540 (58.8%) | 0.0021 | 642 (59.2%) | 626 (57.7%) | 0.030 |
| SAMA; n (%)* | 6 (3.6%) | 7 (4.2%) | -0.0030 | 38 (4.1%) | 42 (4.6%) | -0.0024 | 044 (4.1%) | 049 (4.5%) | -0.020 |
| SABA/SAMA; n (%)* | 6 (3.6%) | 8 (4.8%) | -0.0059 | 52 (5.7%) | 50 (5.4%) | 0.0013 | 058 (5.4%) | 058 (5.4%) | 0.000 |
| ICS; n (%)* | 138 (83.6%) | 137 (83.0%) | 0.0007 | 813 (88.5%) | 805 (87.6%) | 0.0010 | 951 (87.7%) | 942 (86.9%) | 0.024 |
| LABA without formoterol; n (%)* | 2 (1.2%) | 3 (1.8%) | -0.0049 | 31 (3.4%) | 33 (3.6%) | -0.0011 | 033 (3.0%) | 036 (3.3%) | -0.017 |
| LAMA; n (%)* | 16 (9.7%) | 15 (9.1%) | 0.0020 | 106 (11.5%) | 114 (12.4%) | -0.0026 | 122 (11.3%) | 129 (11.9%) | -0.019 |
| LABA/ICS without mometasone-formoterol; n (%)* | 54 (32.7%) | 55 (33.3%) | -0.0010 | 253 (27.5%) | 266 (28.9%) | -0.0026 | 307 (28.3%) | 321 (29.6%) | -0.029 |
| Blood eosinophilia test ; n (%)* | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 3 (0.3%) | 3 (0.3%) | 0.0000 | 003 (0.3%) | 003 (0.3%) | 0.000 |
| Serum immunoglobulin E (IgE) level test; n (%)* | 2 (1.2%) | 2 (1.2%) | 0.0000 | 26 (2.8%) | 33 (3.6%) | -0.0045 | 028 (2.6%) | 035 (3.2%) | -0.036 |
| H2 blocker; n (%)* | 4 (2.4%) | 2 (1.2%) | 0.0089 | 33 (3.6%) | 32 (3.5%) | 0.0005 | 037 (3.4%) | 034 (3.1%) | 0.030 |
| Oxygen codes; n (%)* | 4 (2.4%) | 5 (3.0%) | -0.0037 | 16 (1.7%) | 14 (1.5%) | 0.0003 | 020 (1.8%) | 019 (1.8%) | 0.000 |
| Respiratory arrest/dependence on oxygen; n (%)* | 0 (0.0%) | 1 (0.6%) | -0.0037 | 6 (0.7%) | 6 (0.7%) | 0.0000 | 006 (0.6%) | 007 (0.6%) | 0.000 |
| | (0.070) | 1 (3.070) | 0.0110 | 0 (0.770) | 0 (0.770) | 3.3000 | 333 (3.070) | 55. (0.0/0) | 3.000 |

<sup>\*</sup>Included in the 1:1 PS matching model